Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

| MD Anderson IND | MD Anderson IND Sponsor Cover Sheet |
|---|---|
| Protocol ID | 2015-0948 |
| Protocol Title | Phase II Study for the Evaluation of Efficacy of Pembrolizumab (MK- |
| | 3475) in Patients with Rare Tumors |
| Protocol Phase | Phase II |
| <b>Protocol Version</b> | 17 |
| Version Date | 01/27/2023 |
| Protocol PI | Aung Naing, MD |
| Department | Department Investigational Cancer Therapeutics |
| IND Sponsor | IND Sponsor MD Anderson Cancer Center |
| IND# | 130086 |

Product: MK-3475


## TITLE: Phase II Study for the Evaluation of Efficacy of Pembrolizumab (MK-3475) in Patients with Rare Tumors

PRINCIPAL INVESTIGATOR: Aung Naing, MD

#### SUPPORTER and DRUG SUPPLY:

Merck Sharp & Dohme Corp., a subsidiary of Merck & Co., Inc.

(hereafter referred to as the Supporter or Merck)

One Merck Drive

P.O. Box 100

Whitehouse Station, NJ 08889-0100, U.S.A.

#### **SPONSOR (IND Holder):**

## The University of Texas MD Anderson Cancer Center

(hereafter referred to as the MDACC IND or Sponsor)

Aman Buzdar, M.D.

Vice President for Clinical Research Administration

University of Texas M. D. Anderson Cancer Center

1515 Holcombe Blvd., Unit 1636

Houston, TX 77030

**IND NUMBER:** 130086

## **Protocol Version History:**

Version 00, Dated 11-Dec-2015

Version 01, Dated 04-Jan-2016

Version 02, Dated 06-Jan-2016

Version 03, Dated 19-Jan-2016

Version 04, Dated 12-Feb-2016

Version 05, Dated 13-May-2016

Version 06, Dated 15-Jul-2016

Version 07, Dated 24-Aug-2016

Version 08, Dated 28-Nov-2016

v ci sion 00, Datcu 20-1101-2010

Version 09, Dated 30-Jan-2017

Version 10, Dated 23-Mar-2017

Version 11, Dated 14-Dec-2017

Version 12, Dated 11-Sep-2018

Version 13, Dated 02-Apr-2019

Version 14, Dated 17-Jul-2020

Version 15, Dated 29-Jan-2021

Version 16, Dated 06-Jan-2022

Version 17, Dated 27-Jan-2023

## **TABLE OF CONTENTS**

| 1.0 | TR | SIAL SUMMARY | 8 |
|-----|-------|---------------------------------------------------------|------|
| 2.0 | TR | RIAL DESIGN | . 10 |
| 2. | .1 | Trial Design | . 10 |
| 2. | .2 | Гrial Diagram | . 13 |
| 3.0 | OE | BJECTIVES & HYPOTHESES | . 14 |
| 3. | .1 | Primary Objective | . 14 |
| | 3.1.1 | Secondary Objectives | . 14 |
| | 3.1.2 | Exploratory Objectives: | . 14 |
| 3. | .2 | Hypotheses: | . 15 |
| 4.0 | BA | CKGROUND & RATIONALE | . 15 |
| 4. | .1 | Background | . 15 |
| | 4.1.1 | Pharmaceutical and Therapeutic Background | . 15 |
| | 4.1.2 | Preclinical and Clinical Trial Data | . 16 |
| 4. | .2 | Rationale | . 17 |
| | 4.2.1 | Rationale for the Trial and Selected Subject Population | . 17 |
| | 4.2.2 | Rationale for Dose Selection/Regimen/Modification | . 18 |
| | 4.2.3 | Rationale for Endpoints | . 19 |
| 4. | .3 | Study Updates | . 23 |
| 5.0 | SU | BJECT ELIGIBILITY | . 24 |
| 5. | .1 5 | Study Population | . 24 |
| | 5.1.1 | Diagnosis/Condition for Entry into the Trial | . 24 |
| | 5.1.2 | Subject Inclusion Criteria | . 24 |

Protocol/Amendment No.: Version 17/ MDACC#2015-0948

| 5.1 | .3 Subject Exclusion Criteria | 26 |
|---|---|---|
| 5.2 | Trial Treatments | 28 |
| 5.2 | Dose Selection/Modification | 28 |
| 5.2 | 2.2 Timing of Dose Administration | 34 |
| 5.2 | 2.3 Continuing Study Drug Administration after Initial Evidence of Radiolo Disease Progression | |
| 5.2 | 2.4 Trial Blinding/Masking | 35 |
| 5.3 | Randomization or Treatment Allocation | 35 |
| 5.4 | Stratification | 36 |
| 5.5 | Concomitant Medications/Vaccinations (Allowed & Prohibited) | 36 |
| 5.5 | 7.1 Acceptable Concomitant Medications | 36 |
| 5.5 | 2.2 Prohibited Concomitant Medications | 36 |
| 5.6 | Rescue Medications & Supportive Care | 37 |
| 5.6 | 5.1 Supportive Care Guidelines | 37 |
| 5.7 | Diet/Activity/Other Considerations | 40 |
| 5.7 | '.1 Diet | 40 |
| 5.7 | 7.2 Contraception | 40 |
| 5.7 | '.3 Use in Pregnancy | 41 |
| 5.7 | '.4 Use in Nursing Women | 41 |
| 5.8 | Subject Withdrawal/Discontinuation Criteria | 41 |
| 5.8 | 3.1 Discontinuation of Study Therapy after CR | 43 |
| 5.9 | Subject Replacement Strategy | 43 |
| 5.10 | Clinical Criteria for Early Trial Termination | 43 |
| 6.0 | TRIAL FLOW CHART | <b> 4</b> 4 |
| 6.1 | Study Flow Chart | <b> 4</b> 4 |


| 7.0 | TR | IAL PROCEDURES | . 48 |
|---|---|---|---|
| 7. | 1 7 | Frial Procedures | . 48 |
| | 7.1.1 | Administrative Procedures | . 48 |
| | 7.1.2 | Clinical Procedures/Assessments | . 51 |
| | 7.1.3 | Laboratory Procedures/Assessments | . 60 |
| | 7.1.4 | Other Procedures | . 62 |
| | 7.1.5 | Visit Requirements | . 62 |
| 7. | <b>2</b> A | Assessing and Recording Adverse Events | . 65 |
| | 7.2.1 | Definition of an Overdose for This Protocol and Reporting of Overdose to the IND Sponsor and to Merck | . 66 |
| | 7.2.2 | Reporting of Pregnancy and Lactation to the IND Sponsor and to Merck | . 67 |
| | 7.2.3 | Immediate Reporting of Adverse Events to the IND Sponsor and to Merck | . 67 |
| | 7.2.4 | Evaluating Adverse Events | . 70 |
| | 7.2.5 | Sponsor Responsibility for Reporting Adverse Events | . 73 |
| 8.0 | ST | ATISTICAL ANALYSIS PLAN | . 73 |
| 8. | 1 5 | Statistical Analysis Plan Summary | . 73 |
| | 8.1.1 | General Analyses | . 73 |
| | 8.1.2 | Efficacy Analyses | . 73 |
| | 8.1.3 | Safety Analysis | . 74 |
| | 8.1.4 | Power and Sample Size | . 75 |
| | 8.1.5 | Interim Analyses | . 75 |
| 8. | 2 5 | Statistical Analysis Plan | . 76 |
| | 8.2.1 | Responsibility for Analyses | . 76 |
| 8. | 3 5 | Study Objectives | . 76 |
| | 8.3.1 | Primary Objective | . 76 |


| | 8.3.2 | Secondary Objectives | 76 |
|---|---|---|---|
| | 8.3.3 | Exploratory Objectives: | 76 |
| 8 | 8.4 | Hypotheses: | 77 |
| 8 | 8.5 | Analysis Endpoints | . 77 |
| | 8.5.2 | Analysis Populations | 79 |
| | 8.5.3 | Statistical Methods | 79 |
| 9.0 | | ABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL UPPLIES | |
| 9 | 9.1 | Investigational Product | 80 |
| 9 | 9.2 | Packaging and Labeling Information | 80 |
| 9 | 9.3 | Clinical Supplies Disclosure | 81 |
| 9 | 9.4 | Storage and Handling Requirements | . 81 |
| 9 | 9.5 | Returns and Reconciliation | . 81 |
| 10. | 0 A | DMINISTRATIVE AND REGULATORY DETAILS | . 81 |
| | 10.1 | Confidentiality | . 81 |
| | 10.1. | 1 Confidentiality of Data | 81 |
| | 10.1. | 2 Confidentiality of Subject Records | 82 |
| | 10.1. | 3 Confidentiality of Investigator Information | 82 |
| | 10.1. | 4 Data Sharing | 82 |
| | 10.2 | Compliance with Financial Disclosure Requirements | . 84 |
| | 10.3 | Compliance with Law, Audit and Debarment | . 84 |
| - | 10.4 | Compliance with Trial Registration and Results Posting Requirements | 86 |
| | 10.5 | Quality Management System | 86 |
| | 10.6 | Data Management | 86 |
| 11 | 0 A1 | PPENDICES | 88 |


27Jan2022


## 1.0 TRIAL SUMMARY

| Abbreviated Title | Phase II Pembrolizumab (MK-3475) in Rare Tumors |
|---|---|
| Trial Phase | П |
| Clinical Indication | Subjects will be enrolled into one of the following 10 tumor cohorts: 1) Squamous cell carcinoma of the skin 2) Small cell malignancies of non-pulmonary origin 3) Adrenocortical carcinoma 4) Medullary renal cell carcinoma 5) Carcinoma of unknown primary 6) Penile carcinoma 7) Vascular sarcoma 8) Germ Cell Tumor 9) Paraganglioma-pheochromocytoma 10) Other rare tumor histologies |
| Trial Type | Interventional |
| Type of control | No Treatment Control |
| Route of administration | Intravenous |
| Trial Blinding | Unblinded, Open-Label |
| Treatment Groups | Pembrolizumab (MK-3475) 200 milligrams intravenous infusion every 3 weeks |
| Number of trial subjects | 250 Subjects |
| Estimated enrollment period | March 2016-December 2021 |
| Estimated duration of trial | The investigator estimates that the trial will require approximately 24 months from the time the first subject signs the informed consent until the last subject's last visit |
| Duration of Participation | Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final protocol-specified contact. After a screening phase of 28 days, eligible subjects will receive treatment on Day 1 of each 21 day dosing cycle. Treatment with pembrolizumab (MK-3475) will continue until documented confirmed radiological disease progression or clinical progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements; subject receives 24 months of study medication, or administrative reasons. Subjects who attain a complete response may consider stopping trial treatment if they meet criteria for holding therapy. Subjects who stop trial treatment after receiving 24 months of study medication for reasons other than disease progression or intolerability or who attain a complete response and stop trial treatment may be eligible for up to one year of retreatment after experiencing disease progression. The decision to retreat will be at the discretion of the investigator only if they meet the criteria for retreatment and the trial is ongoing. After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (study drug-related serious adverse events will be collected for 90 days after the end of treatment). Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, |


| withdrawing consent, or becoming lost to follow-up. Investigators will |
|------------------------------------------------------------------------|
| collect survival data for patients after progression of disease unless |
| patient fully withdrew consent to participate in the study using |
| information from a chart review, patient visit, or telephone call. |

Product: MK-3475


10

## 2.0 TRIAL DESIGN

## 2.1 Trial Design

This is a single-center, open-label, phase II trial of pembrolizumab (MK-3475) in patients with and without programmed death-ligand 1 (PD-L1) positive advanced tumors to be conducted at the University of Texas MD Anderson Cancer Center.

Participation in this trial will be dependent upon pathology or histologic confirmation of an advanced tumor type. Subjects will be enrolled into one of the following 10 tumor cohorts:

- 1) Squamous cell carcinoma of the skin
- 2) Small cell malignancies of non-pulmonary origin
- 3) Adrenocortical carcinoma
- 4) Medullary renal cell carcinoma
- 5) Carcinoma of unknown primary
- 6) Penile carcinoma
- 7) Vascular sarcoma
- 8) Germ Cell Tumor
- 9) Paraganglioma-pheochromocytoma
- 10) Other rare tumor histologies.

In Cohort 10, "Other rare tumor histologies," the following tumor types will be excluded: melanoma, non-small cell lung cancer, hepatocellular carcinoma, Merkel cell carcinoma, colon or rectal adenocarcinoma, anal canal squamous cell carcinoma, pancreas adenocarcinoma, esophageal squamous cell carcinoma or adenocarcinoma (including GE junction), biliary tract adenocarcinoma (gallbladder and biliary tree but excluding ampulla of vater cancers), carcinoid tumors, neuroendocrine carcinomas (well or moderately differentiated pancreatic neuroendocrine tumor), ER-positive HER2-negative breast cancer, triple negative breast cancer, ovarian epithelial, fallopian tube or primary peritoneal carcinoma, endometrial carcinoma, cervical squamous cell cancer, vulvar squamous cell carcinoma, small cell lung cancer, malignant pleural mesothelioma, thyroid cancer (papillary or follicular subtype), glioblastoma gland carcinoma, nasopharyngeal carcinoma, leiomyosarcoma, prostate adenocarcinoma, gastric adenocarcinoma, and small bowel malignancy.

Patients will be enrolled regardless of their PD-L1 expression status. Patients will supply tissue from an archival tissue sample or newly obtained biopsy (if archival tissue is not available) of a tumor lesion not previously irradiated (tumors progressing in a prior site of radiation are allowed for PD-L1 characterization, other exceptions may be considered after PI consultation). This specimen will be evaluated at a central laboratory for expression status of PD-L1 by immunohistochemistry (IHC).

Toxicities will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Subjects will be evaluated every 3 cycles

Product: MK-3475

11 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

= every 9 weeks (63 days  $\pm$ 7 days) with radiographic imaging to assess response to treatment. After 6 months, at the physician's discretion, if patients have had complete response (CR), partial response (PR) or stable disease (SD) > 27 weeks, then radiographic imaging may be performed every 12 weeks (4 cycles or 84 days  $\pm$  7 days). Response Evaluation Criteria in Solid Tumors (RECIST) 1.11 or immune-related RECIST (irRECIST) or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated will be used as the primary and secondary efficacy endpoint of response rate.

Treatment with pembrolizumab (MK-3475) will continue until documented radiological disease progression or clinical progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, completion of 24 months of treatment with pembrolizumab (MK-3475), or administrative reasons. Subjects who attain an investigatordetermined confirmed complete response (CR) may consider stopping trial treatment after receiving at least 27 weeks (9 cycles) of treatment. In addition, subjects who discontinue after at least 24 months of therapy for reasons other than disease progression or intolerability, or who discontinue after attaining a CR and had at least 2 treatments beyond initial CR, may be eligible for up to one year of retreatment if they subsequently experience radiographic disease progression. The decision to retreat will be at the discretion of the investigator only if no cancer treatment was administered since the last dose of pembrolizumab (MK-3475), the subject still meets the safety parameters listed in the Inclusion/Exclusion criteria and the trial remains open. After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (study drug-related serious adverse events will be collected for 90 days after the end of treatment). Subjects who discontinue treatment for reasons other than disease progression will have post-treatment follow-up of disease status until disease progression, or initiating a non-study cancer treatment, or withdrawing consent, or becoming lost to follow-up. Investigators will collect survival data for patients after progression of disease unless patient fully withdrew consent to participate in the study using information from a chart review, patient visit, or telephone call. The telephone call will be less than five minutes to obtain information regarding survival status.

Immunotherapeutic agents such as pembrolizumab (MK-3475) may produce antitumor effects by potentiating endogenous cancer-specific immune responses. The response patterns seen with such an approach may extend beyond the typical time course of responses seen with cytotoxic agents, and can manifest as a clinical response after an initial increase in tumor burden or even the appearance of new lesions. If initial radiologic imaging shows progressive disease (PD), tumor assessment should be repeated  $\geq 4$  weeks later in order to confirm PD with the option of continuing treatment per below while awaiting radiologic confirmation of progression. If repeat imaging shows a reduction in the tumor burden compared to the initial scan demonstrating PD, treatment may be continued as per treatment calendar. If repeat imaging confirms progressive disease, subjects will be discontinued from study therapy. In determining whether or not the tumor burden has increased or decreased, Investigators should consider all target lesions as well as non-target lesions.

Product: MK-3475 12 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

The primary objective of the trial is to evaluate efficacy by evaluation of non-progression rate (NPR) at 27 weeks (9 cycles) as defined as the percentage of patients who are alive and progression-free at 27 weeks (9 cycles) as assessed by RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated, of pembrolizumab (MK-3475) in subjects with or without PD-L1 positive advanced tumors. Secondary objectives include evaluating safety and tolerability of pembrolizumab (MK-3475); correlating efficacy, non-progression rate (NPR) at 27 weeks (9 cycles), objective response (CR or PR), clinical benefit (CR, PR, or stable disease [SD] >/=4 months), progression-free survival (PFS), overall survival (OS) and duration of response (DOR) to PD-L1 status; and identifying imaging characteristics associated with immunological changes in tumor following treatment with pembrolizumab.

Product: MK-3475
27Jan2022

## 2.2 Trial Diagram

The trial design is depicted in Figure 1.



Figure 1: Dosing and Correlative Schema

Patients may be co-enrolled on other protocols in which the PBMC and tissue samples will be utilized for analyses.

Product: MK-3475

Product: MK-3475
27Jan2022

#### 3.0 OBJECTIVES & HYPOTHESES

## 3.1 Primary Objective

**Objective**: To obtain early indication of efficacy by evaluation of non-progression rate (NPR) at 27 weeks as defined as the percentage of patients who are alive and progression-free at 27 weeks as assessed by RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated in patients with advanced tumor types receiving pembrolizumab.

## 3.1.1 Secondary Objectives

- (1) **Objective**: To correlate efficacy by evaluation of tumor size to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.
- (2) **Objective:** To evaluate safety and tolerability of pembrolizumab in patients with advanced tumors.
- (3) **Objective:** To evaluate the percentage of patients with objective response (CR or PR), clinical benefit (CR, PR, or stable disease [SD] >/=4 months), progression free survival (PFS), overall survival (OS), and duration of response (DOR) as assessed by RECIST v1.1 in patients with advanced tumor types receiving pembrolizumab.
- (4) **Objective:** To evaluate the percentage of patients with objective response (CR or PR), clinical benefit (CR, PR, or SD >/=4 months), PFS, and DOR as assessed by irRECIST in patients with advanced tumor types receiving pembrolizumab.
- (5) **Objective:** To correlate the NPR at 27 weeks (9 cycles), objective response (CR or PR), clinical benefit (CR, PR, or SD >/=4 months), PFS, OS, and DOR to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.

## 3.1.2 Exploratory Objectives:

- (1) **Objective:** To evaluate the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness in patients with advanced tumor types receiving pembrolizumab.
- (2) **Objective:** To correlate the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.
- (3) **Objective:** To identify imaging characteristics associated with immunological changes in tumor following treatment with pembrolizumab.

Product: MK-3475

15 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

(4) Objective: To compare tumor mutation burden and serial assessment of mutation status in biopsies obtained at baseline and progression in patients with advanced tumor types receiving pembrolizumab.

- (5) **Objective:** To evaluate patient-reported outcomes (PRO) utilizing the National Cancer Institute (NCI) Patient-Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) questionnaires.
- (6) **Objective:** For patients that experience dermatologic irAEs, to compare the skin microbiome of normal (non-rash) skin to skin microbiome of area with rash.
- (7) **Objective:** For patients that experience oral irAEs, to assess the oral microbiome at baseline, at onset of toxicity, and time of tumor restaging
- (8) Objective: For patients that experience gut irAEs, to assess the gut microbiome at baseline, onset of toxicity, time of tumor restaging, and End of Treatment visit per the parent treatment protocol.
- (9) Objective: To analyze tumor-infiltrating lymphocytes using H&E (hematoxylin and eosin) stained whole slide images.

#### 3.2 **Hypotheses:**

Intravenous administration of single agent pembrolizumab (MK-3475) to subjects with a given PD-L1 positive advanced tumor type will result in an NPR at 27 weeks (9 cycles) greater than 20% based on RECIST v1.1 or irRECIST criteria or according to tumor evaluation criteria best suitable and accepted for the tumor type evaluated.

#### 4.0 BACKGROUND & RATIONALE

#### **Background** 4.1

Refer to the Investigator's Brochure (IB)/approved labeling for detailed background information on pembrolizumab (MK-3475).<sup>2</sup>

## 4.1.1 Pharmaceutical and Therapeutic Background

The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+

Product: MK-3475


16

effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in many solid tumors.

The programmed death 1 (PD-1) receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4 which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2). The structure of murine PD-1 has been resolved. PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail which is responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosinebased switch motif (ITSM). Following T-cell stimulation, PD-1 recruits the tyrosine phosphatases SHP-1 and SHP-2 to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ and ZAP70 which are involved in the CD3 T-cell signaling cascade. The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from that of CTLA-4 as both molecules regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, T regs and Natural Killer cells. Expression has also been shown during thymic development on CD4-CD8- (double negative) T-cells as well as subsets of macrophages and dendritic cells. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types, including non-hematopoietic tissues as well as in various tumors. Both ligands are type I transmembrane receptors containing both IgV- and IgC-like domains in the extracellular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium, whereas PD-L2 protein is only detectably expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PD-L1 serves to dampen unwarranted T-cell function in peripheral tissues. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. PD-1 has been suggested to regulate tumor-specific T-cell expansion in subjects with melanoma (MEL). This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

#### 4.1.2 Preclinical and Clinical Trial Data

Refer to the Investigator's Brochure for Preclinical and Clinical data.<sup>2</sup>

Product: MK-3475

17 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

#### 4.2 Rationale

## 4.2.1 Rationale for the Trial and Selected Subject Population

Intact immune surveillance plays a significant role in controlling development of neoplastic transformation.<sup>3</sup> PD-1 is an immune-checkpoint receptor expressed by T cells. PD-L1 is expressed in the tumor microenvironment of various cancers. Upon binding to either of its ligands, PD-L1 or PD-L2, the PD-1 pathway negatively regulates T-cell effector functions. Increased expression of PD-L1 and an immunosuppressive microenvironment are associated with ineffective host immune response and subsequent disease progression in multiple tumor malignancies. There is a strong correlation between presence of effective lymphocytes and favorable prognosis in different types of malignancies.<sup>4-6</sup> Tumors take advantage of immune check points such as the PD-1/PD-L1 pathway to evade immune destruction, resulting in disease progression.<sup>7,8</sup> To overcome tumor immune suppression and to establish an effective antitumor immune response, it is necessary to overcome multiple immunosuppressive mechanisms.<sup>9,10</sup> Anti-PD1, anti-PD-L1, and anti-CTLA-4 are designed to block immune checkpoints. These checkpoint inhibitors thereby decrease immune suppression and increase the antitumor effect.

Pembrolizumab (also known as lambrolizumab and previously known as MK-3475) is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. The t1/2 of pembrolizumab is approximately 2-3 weeks (14-21 days), and with no indication of dose dependency of half-life among three dose groups (1, 3, and 10 mg/kg), which supports a dosing interval of every 2 or 3 weeks. 11 Steady-state trough concentrations were 20% greater in patients receiving 10 mg/kg every 2 weeks than in those receiving the same dose every 3 weeks. Pembrolizumab has shown overall response rates of approximately 38% in patients with melanoma and  $\sim 20\%$  in patients with non-small cell lung cancer. In September 2014, the FDA granted early approval for pembrolizumab in melanoma patients with BRAF V600 mutation following ipilimumab therapy. 12

Currently, a single agent pembrolizumab trial is being conducted in over 20 PD-L1 expressing tumors including: colon or rectal adenocarcinoma, anal canal squamous cell carcinoma, pancreas adenocarcinoma, esophageal squamous cell carcinoma, adenocarcinoma (including GE junction), biliary tract adenocarcinoma (gallbladder and biliary tree but excluding ampulla of vater cancers), carcinoid tumors, neuroendocrine carcinomas (well or moderately differentiated pancreatic neuroendocrine tumor), ER+/HER2-negative breast cancer, ovarian epithelial, fallopian tube or primary peritoneal carcinoma, endometrial carcinoma, cervical squamous cell cancer, vulvar squamous cell carcinoma, small cell lung cancer, mesothelioma (malignant pleural mesothelioma), thyroid cancer (papillary or follicular subtype), salivary gland carcinoma, nasopharyngeal carcinoma, glioblastoma multiforme, leiomyosarcoma, prostate adenocarcinoma (NCT02054806).

Progress is unfolding in the understanding of how the immune system can modulate tumor progression or effective responses against cancer.<sup>13</sup> In some studies, the levels of PD-L1

Product: MK-3475

18 27Jan2022 Protocol/Amendment No.: Version 17/ MDACC#2015-0948

expression have correlated with clinical outcome. 14-16 However, the prognostic impact of PD-L1 expression still needs to be defined in rare tumor types.

Our strategy for this study is to focus on advanced rare types with and without PD-L1expressing tumors. We will exclude all types of tumors that are enrolled in the current Phase 1B study of MK-3475-028 (NCT02054806). In this study, our goal is to characterize the presence of PD-L1 expression in advanced tumor tissues and to correlate levels of PD-L1 expression with clinico-pathological features as well as survival outcomes.

## 4.2.2 Rationale for Dose Selection/Regimen/Modification

An open-label Phase I trial (Protocol 001) is being conducted to evaluate the safety and clinical activity of single agent MK-3475. The dose escalation portion of this trial evaluated three dose levels, 1 mg/kg, 3 mg/kg, and 10 mg/kg, administered every 2 weeks (Q2W) in subjects with advanced solid tumors. All three dose levels were well tolerated and no dose-limiting toxicities were observed. This first in human study of MK-3475 showed evidence of target engagement and objective evidence of tumor size reduction at all dose levels (1 mg/kg, 3 mg/kg and 10 mg/kg Q2W). No MTD has been identified to date. 10.0 mg/kg Q2W, the highest dose tested in PN001, will be the dose and schedule utilized in Cohorts A, B, C and D of this protocol to test for initial tumor activity. Recent data from other clinical studies within the MK-3475 program has shown that a lower dose of MK-3475 and a less frequent schedule may be sufficient for target engagement and clinical activity.

PK data analysis of MK-3475 administered Q2W and Q3W showed slow systemic clearance, limited volume of distribution, and a long half-life.<sup>2</sup> Pharmacodynamic data (IL-2 release assay) suggested that peripheral target engagement is durable (>21 days). This early PK and pharmacodynamic data provides scientific rationale for testing a Q2W and Q3W dosing schedule.

A population pharmacokinetic analysis has been performed using serum concentration time data from 476 patients. Within the resulting population PK model, clearance and volume parameters of MK-3475 were found to be dependent on body weight. The relationship between clearance and body weight, with an allometric exponent of 0.59, is within the range observed for other antibodies and would support both body weight normalized dosing or a fixed dose across all body weights. MK-3475 has been found to have a wide therapeutic range based on the melanoma indication. The differences in exposure for a 200 mg fixed dose regimen relative to a 2 mg/kg Q3W body weight based regimen are anticipated to remain well within the established exposure margins of 0.5 - 5.0 for MK-3475 in the melanoma indication. The exposure margins are based on the notion of similar efficacy and safety in melanoma at 10 mg/kg Q3W vs. the proposed dose regimen of 2 mg/kg Q3W (i.e. 5-fold higher dose and exposure). The population PK evaluation revealed that there was no significant impact of tumor burden on exposure. In addition, exposure was similar between the NSCLC and melanoma indications. Therefore, there are no anticipated changes in exposure between different indication settings.

Product: MK-3475


19

The rationale for further exploration of 2 mg/kg and comparable doses of pembrolizumab in solid tumors is based on: 1) similar efficacy and safety of pembrolizumab when dosed at either 2 mg/kg or 10 mg/kg Q3W in melanoma patients, 2) the flat exposure-response relationships of pembrolizumab for both efficacy and safety in the dose ranges of 2 mg/kg Q3W to 10 mg/kg Q3W, 3) the lack of effect of tumor burden or indication on distribution behavior of pembrolizumab (as assessed by the population PK model) and 4) the assumption that the dynamics of pembrolizumab target engagement will not vary meaningfully with tumor type.

The choice of the 200 mg Q3W as an appropriate dose for the switch to fixed dosing is based on simulations performed using the population PK model of pembrolizumab showing that the fixed dose of 200 mg every 3 weeks will provide exposures that 1) are optimally consistent with those obtained with the 2 mg/kg dose every 3 weeks, 2) will maintain individual patient exposures in the exposure range established in melanoma as associated with maximal efficacy response and 3) will maintain individual patients exposure in the exposure range established in melanoma that are well tolerated and safe.

A fixed dose regimen will simplify the dosing regimen to be more convenient for physicians and to reduce potential for dosing errors. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities and reduce wastage.

## 4.2.3 Rationale for Endpoints

## 4.2.3.1 Efficacy Endpoints

The primary objective of this study is to evaluate the efficacy by evaluation of non-progression rate (NPR) at 27 weeks as defined as the percentage of patients who are alive and progression-free at 27 weeks as assessed by RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated, of pembrolizumab (MK-3475) in subjects with and without PD-L1 positive advanced tumors. Response rates per RECIST v1.1 or irRECIST will be evaluated. The same method of assessment used to characterize each identified and reported lesion at baseline must be used in all subsequent imaging assessments. Response assessments determined by irRECIST will be compared with those of derived using RECIST v1.1.

RECIST v1.1 or irRECIST will be adapted to account for the unique tumor response characteristics seen with treatment of pembrolizumab (MK-3475). Immunotherapeutic agents such as pembrolizumab (MK-3475) may produce antitumor effects by potentiating endogenous cancer-specific immune responses. The response patterns seen with such an approach may extend beyond the typical time course of responses seen with cytotoxic agents, and can manifest a clinical response after an initial increase in tumor burden or even the appearance of new lesions. Standard RECIST may not provide an accurate response assessment of immunotherapeutic agents such as pembrolizumab (MK-3475). Therefore, RECIST v1.1 will be used with the following adaptations:

• If radiologic imaging shows initial PD, tumor assessment should be repeated ≥4

Product: MK-3475

20 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

weeks later in order to confirm PD with the option of continuing treatment per below while awaiting radiologic confirmation of progression. If repeat imaging shows a reduction in the tumor burden compared to the initial scan demonstrating PD, treatment may be continued / resumed. If repeat imaging confirms progressive disease, subjects will be discontinued from study therapy (exception noted in Section 7.1.2.6). In determining whether or not the tumor burden has increased or decreased, investigators should consider all target lesions as well as non-target lesions.

In subjects who have initial evidence of radiological PD, it is at the discretion of the treating physician whether to continue a subject on study treatment until repeat imaging is obtained a minimum of 4 weeks later. This clinical judgment decision should be based on the subject's overall clinical condition, including performance status, clinical symptoms, and laboratory data. Subjects may receive pembrolizumab (MK-3475) treatment while waiting for confirmation of PD if they are clinically stable as defined by the following criteria:

- Absence of signs and symptoms indicating disease progression
- No decline in ECOG performance status
- Absence of rapid progression of disease
- Absence of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention.

When feasible, subjects should not be discontinued until progression is confirmed. This allowance to continue treatment despite initial radiologic progression takes into account the observation that some subjects can have a transient tumor flare in the first few months after the start of immunotherapy, but with subsequent disease response. Subjects that are deemed clinically unstable are not required to have repeat imaging for confirmation of progressive disease.

## 4.2.3.2 Safety Endpoints

The secondary safety objective of this study is to characterize the safety and tolerability of pembrolizumab (MK-3475) in subjects with or without PD-L1 positive advanced tumors. The safety analysis will be based on subjects who experienced toxicities as defined by CTCAE criteria. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received pembrolizumab (MK-3475), including serious adverse events (SAEs) and events of clinical interest (ECIs).

Safety will be assessed by reported adverse experiences using CTCAE, Version 4.03. The attribution to drug, time-of-onset, duration of the event, its resolution, and any concomitant medications administered will be recorded. AEs will be analyzed including but not limited to all AEs, SAEs, fatal AEs, and laboratory changes. Furthermore, specific immune-related adverse events (irAEs) will be collected and designated as immune-related events of clinical interest (ECIs) as described in Section 7.2.3.2.

Product: MK-3475

21 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

Patients enrolled on this study will be approached for co-enrollment on PA15-0315 prospective study to assess immune-related adverse events when receiving immunotherapy at the University of Texas MD Anderson Cancer Center (Aung Naing, MD). All samples and scans will be collected using procedures characterized in this protocol, and all patients will be consented for procedures done under this optional protocol separately.

#### 4.2.3.3 Biomarker Research

Additional biomarker research to identify factors important for pembrolizumab (MK-3475) therapy will also be pursued. For example, tumor and blood samples from this study may undergo proteomic, genomic and transcriptional analyses. Additional research may evaluate factors important for predicting responsiveness or resistance to pembrolizumab (MK-3475) therapy and other immunologic targets.

Participation in this trial will be dependent upon supplying tissue from an archival tissue sample or newly obtained biopsy (if archival tissue is not available) of a tumor lesion not previously irradiated (tumors progressing in a prior site of radiation are allowed for PD-L1 characterization, other exceptions may be considered after PI consultation). This specimen will be evaluated at a central laboratory for expression status of PD-L1 by immunohistochemistry (IHC). Baseline, on-treatment and time of progression (if patients have had CR/PR/or SD for > 27 weeks) biopsies will be obtained for evaluation of the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness. Biopsies will be performed provided that there is technically biopsiable tumor, and it is safe for patient to undergo biopsy. In Cohort 9: Paraganglioma-pheochromocytoma or Cohort 10, where there is prominent bony disease, biopsies may not be possible due to the nature of the disease.

Peripheral blood mononuclear cell (PBMC) will be collected at baseline, tumor restaging, in conjunction with biopsies, and time of progression (if patients have had CR/PR/or SD for > 27 weeks). These samples will be analyzed for the NanoString assay that will evaluate immunerelated gene expression signatures and the potential to predict benefit from pembrolizumab.

Patients enrolled in this study will be approached for co-enrollment on PA11-0852 Clearinghouse protocol at the University of Texas MD Anderson Cancer Center (Funda Meric-Bernstam, MD) to assess tumor mutation burden and genomic alterations detected in cfDNA. As per the PA11-0852 Clearinghouse protocol, the optional tumor biopsies from baseline and the time of progression (if progression after response or unexpected rapid progression), and serial plasma samples will be analyzed. Development of new mutations or reversal of the mutations will be analyzed and correlated with clinical response. This will be our exploratory objective and no formal statistical analysis will be done.

## 4.2.3.4 Patient-Reported Outcomes

In collaboration with the Department of Symptom Research, we will use pre-specified selected items from the National Cancer Institute (NCI) Patient-Reported Outcomes version 1.0 of the

Product: MK-3475


22

Common Terminology Criteria for Adverse Events (PRO-CTCAE) library of items. The NCI PRO-CTCAE provides a systematic yet flexible tool for descriptive reporting of symptomatic treatment side effects in cancer clinical trials.

Capturing symptomatic toxicity is challenging since the onset and character of adverse events varies within and across trials based on the distinct, on- and off-target toxicity profile of a specific therapy. Thus the approach to measuring symptomatic toxicity must be flexible within and across studies.

The National Cancer Institute's PRO-CTCAE measurement system was developed as a companion to the CTCAE, the standard lexicon for adverse event reporting in cancer trials. It is not intended to be used as a stand alone patient-reported outcome.

The PRO-CTCAE measurement system includes an item library of 124 discrete items representing 78 symptomatic toxicities drawn from the CTCAE. It provides a systematic yet flexible approach to capture symptomatic treatment side effects in trials of new cancer therapies.

For this study, the 20 symptomatic toxicities including oral (dry mouth), gastrointestinal (decreased appetite, nausea, diarrhea, and abdominal pain), respiratory (shortness of breath), cardio/circulatory (swelling), cutaneous (rash, skin dryness, and itchiness), visual/perception (blurred vision), pain (generalized pain, headache, muscle pain, joint pain), sleep/wake (fatigue), sexual (decreased libido), and miscellaneous (chills, increased sweating, and hot flashes) will be used.

PRO-CTCAE responses will be rated using a one-week recall period on a 4-point scale, with 0="Never" or "Never" and 4="Very severe" or "Very much" or "Almost constantly." PRO-CTCAE responses are scored from 0 to 4, and there are no standardized scoring rules yet established for how to combine attributes into a single score or how best to analyze PRO-CTCAE data longitudinally. PRO-CTCAE scores for each attribute (frequency, severity and/or interference) should be presented descriptively (e.g. summary statistics or graphical presentations). The proportion of missing PRO-CTCAE data should also be summarized to aid interpretation.

We will rely on well-established electronic data-capture methods for the PRO-CTCAE. Depending on patient preference, the PRO-CTCAE can be delivered by a computerized, telephone-based interactive voice response (IVR) system at the patient's preferred time and days of the week or electronically through web-based platforms.

The purpose of this project is to estimate the incidence of treatment-emergent irAEs and conduct serial PRO assessments. We will evaluate how these patients were managed and investigate the outcome. By utilizing the PRO-CTCAE questionnaires, we will examine the relationships of longitudinal patient-reported symptoms with disease progression and clinical outcomes of severe irAEs on patients treated with immunotherapy. These results will provide information that is imperative to providing the most effective patient care.

Product: MK-3475


23

## 4.3 Study Updates

As of Protocol Version 14, cohorts of this study were closed due to lack of efficacy or difficulty in accrual.

- Cohort 2: Small cell malignancies of non-pulmonary origin;
- Cohort 4: Medullary renal cell carcinoma;
- Cohort 6: Penile carcinoma;
- Cohort 8: Germ cell tumor.

In summary, Cohort 2 Small cell malignancies of non-pulmonary origin was closed after 12 patients were treated and none were alive and progression-free at 27 weeks (primary-endpoint of the study) (June 2019).

Cohort 4 Medullary renal cell carcinoma was closed after 5 patients were treated and none were alive and progression-free at 27 weeks (primary-endpoint of the study) (April 2019).

Cohort 6 Penile carcinoma was closed after 3 patients were treated (August 2019). Cohort 6 was difficult to accrue due to eligibility, and 2 of the 3 patients progressed rapidly within 2 months of treatment.

Cohort 8 Germ cell tumor was closed after 12 patients were treated (June 2018). Only 1 patient was alive and progression free at 27 weeks (primary-endpoint of the study).

Product: MK-3475

Product: MK-3475 24 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

#### 5.0 SUBJECT ELIGIBILITY

## 5.1 Study Population

## 5.1.1 Diagnosis/Condition for Entry into the Trial

Male and female subjects with or without PD-L1 positive advanced tumor (as specified in Section 5.1.2) of at least 18 years will be enrolled in this trial.

## 5.1.2 Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

- 1. Be willing and able to provide written informed consent/assent for the trial.
- 2. Be  $\geq$  18 years of age on day of signing informed consent.
- 3. Have measurable disease based on RECIST 1.1 or irRECIST. Only Cohort 9 and Cohort 10 can have evaluable disease (non-measureable lesions). Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Patients may have bone metastatic disease evaluable according to tumor evaluation criteria best suitable and accepted for the tumor type evaluated.
- 4. Have one of the following advanced (unresectable and/or metastatic) solid tumor indications, that has progressed following standard therapies, where standard therapies are available:
  - Squamous cell carcinoma of the skin
  - Adrenocortical carcinoma
  - Carcinoma of unknown primary
  - Vascular sarcoma
  - Paraganglioma-pheochromocytoma
  - Other rare tumor histologies (except those tumor types listed in 5.1.3.)
- 5. Have failed prior treatment within 6 months of consent date.
- 6. Have biopsiable disease. Subjects must have at least one lesion amenable to biopsy. Tumor lesions used for biopsy should not be lesions used as target lesions for response evaluation. In Cohort 9: Paraganglioma-pheochromocytoma or Cohort 10, where there is prominent bony disease, biopsies may not be possible due to the nature of the disease.
- 7. Be willing to provide archival tissue. If archival tissue is not available, a newly obtained core or excisional biopsy of a tumor lesion will be obtained. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day

Product: MK-3475


25
27Jan2022

1. In Cohort 9: Paraganglioma-pheochromocytoma or Cohort 10, where there is prominent bony disease, biopsies may not be possible due to the nature of the disease.

- 8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
- 9. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 28 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values

| System | Laboratory Value |
|---|---|
| Hematological | |
| Absolute neutrophil count (ANC) | ≥1,000 /mcL |
| Platelets | ≥75,000 / mcL |
| Hemoglobin | ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) |
| Renal | |
| Serum creatinine <u>OR</u><br>Measured or calculated <sup>a</sup> creatinine | ≤1.5 X upper limit of normal (ULN) <u>OR</u> |
| clearance | $\geq$ 60 mL/min for subject with creatinine levels $> 1.5 \text{ X}$ |
| (GFR can also be used in place of creatinine or CrCl) | institutional ULN |
| Hepatic | |
| Serum total bilirubin | ≤ 1.5 X ULN <u>OR</u> |
| | Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN |
| AST (SGOT) and ALT (SGPT) | ≤ 2.5 X ULN <u>OR</u><br>≤ 5 X ULN for subjects with liver metastases |
| Albumin | ≥2.5 mg/dL |
| Coagulation | .= |
| International Normalized Ratio (INR) or Prothrombin Time (PT) | ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants |
| Activated Partial Thromboplastin Time (aPTT) | ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants |
| <sup>a</sup> Creatinine clearance should be calculated per institutional standard. | |

- 10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
- 11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Product: MK-3475 26 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

13. For subjects in Cohort 2 (Small cell malignancies of non-pulmonary origin), confirmation of no brain metastases via imaging.

## 5.1.3 Subject Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

- 1. Is currently participating and receiving study therapy or concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment at the time of administration of first dose of trial treatment. Continuation of hormone replacement therapy is permitted. Stable regimens of hormonal therapy i.e. for prostate cancer (e.g. leuprolide, a GnRH agonist), ovarian, or breast cancer are not exclusionary.
- 2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
- 3. Has a known history of active TB (Bacillus Tuberculosis).
- 4. Hypersensitivity to pembrolizumab or any of its excipients.
- 5. Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
  - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  - Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
- 6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and diseases for which the treatment could reasonably include Pembrolizumab and are not part of the excluded tumor type list or not eligible for the phase I trial.
- 7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using

Product: MK-3475


steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

27

- 8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of Pembrolizumab. Note: corticosteroids given within 24 hours of an imaging study for purposes of premedication in patients with hypersensitivity to radiologic contrast agents are allowed.
- 9. Has known history of, or any evidence of active, non-infectious pneumonitis.
- 10. Has an active infection requiring systemic therapy.
- 11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
- 14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
- 15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
- 16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
- 17. Has received a live vaccine within 30 days of planned start of study therapy.
  - Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
- 18. Is participating in Cohort 10 and has melanoma; non-small cell lung cancer; hepatocellular carcinoma; Merkel cell carcinoma; colon or rectal adenocarcinoma; anal canal squamous cell carcinoma; pancreas adenocarcinoma; esophageal squamous cell carcinoma or adenocarcinoma (including GE junction); biliary tract adenocarcinoma (gallbladder and biliary tree but excluding ampulla of vater cancers); carcinoid tumors;

Product: MK-3475


28

neuroendocrine carcinomas (well or moderately differentiated pancreatic neuroendocrine tumor); ER-positive HER2-negative breast cancer; triple negative breast cancer; ovarian epithelial, fallopian tube or primary peritoneal carcinoma; endometrial carcinoma; cervical squamous cell cancer; vulvar squamous cell carcinoma; small cell lung cancer; mesothelioma (malignant pleural mesothelioma); thyroid cancer (papillary or follicular subtype); salivary gland carcinoma; nasopharyngeal carcinoma; glioblastoma multiforme; leiomyosarcoma; prostate adenocarcinoma; gastric adenocarcinoma; or small bowel malignancy.

#### **5.2** Trial Treatments

The treatment to be used in this trial is outlined below in Table 2. One treatment cycle consists of 3 weeks (21 days) of treatment. Pembrolizumab will be given via intravenous (IV) infusion on Day 1 of every cycle. Patients will be restaged at the end of every three cycles (9 weeks). Patients may be allowed to continue treatment after restaging if there is continued clinical response or disease stabilization and patients do not have significant toxicities.

Table 2 Trial Treatment

| Drug | Dose/Potency | Dose<br>Frequency | Route of Administration | Regimen/Treatment<br>Period | Use |
|---|---|---|---|---|---|
| Pembrolizumab (MK-3475) | 200 mg | Q3W | IV Infusion | Day 1 of each 21-<br>Day Cycle | Experimental |
| The pembrolizumab (MK-3475) dosing interval may be withheld due to toxicity as described in Section 5.2.1.2. | | | | | |

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of trial treatments in accordance with the protocol and any applicable laws and regulations.

#### **5.2.1** Dose Selection/Modification

#### **5.2.1.1** Dose Selection

The rationale for selection of doses to be used in this trial is provided in <u>Section 4.0</u> – Background and Rationale.

Details on preparation and administration of pembrolizumab (MK-3475) are provided in the Pharmacy Manual.

#### **5.2.1.2** Dose Modification

Adverse events (both non-serious and serious) associated with pembrolizumab exposure may represent an immunologic etiology. These adverse events may occur shortly after the first dose or several months after the last dose of treatment. Pembrolizumab must be withheld for drug-

Product: MK-3475 29 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

related toxicities and severe or life-threatening AEs as per Table 3 below. See <u>Section 5.6.1</u> for supportive care guidelines, including use of corticosteroids.

For subjects whose dose was withheld due to toxicity, subjects may resume pembrolizumab (MK-3475) upon resolution of toxicity to Grade 0-1 or baseline. This dose would be considered Day 1 of the next cycle and should be in alignment with the new schedule.

Product: MK-3475
27Jan2022

**Table 3 Dose Modification Guidelines for Drug-Related Adverse Events** 

#### **General Instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤10 mg prednisone or equivalent per day within 12 weeks.
- **3.** For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with corticosteroid and/or other therapies | Monitor and follow-up | |
|---|---|---|---|---|---|
| Pneumonitis | Grade 2 | Withhold | Administer corticosteroids (initial dose of 1-2 mg/kg prednisone or equivalent) followed by taper | dose of 1-2 mg/kg prednisone or equivalent) followed by taper symptoms of pneum equivalent followed by taper Evaluate participants | symptoms of pneumonitis • Evaluate participants with suspected |
| | Grade 3 or 4, or recurrent Grade 2 | Permanently discontinue | | <ul> <li>pneumonitis with radiographic imaging and initiate corticosteroid treatment</li> <li>Add prophylactic antibiotics for opportunistic infections</li> </ul> | |
| Diarrhea / Colitis | Grade 2 or 3 | Withhold | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | <ul> <li>Monitor participants for signs and symptoms of enterocolitis (ie, diarrhea, abdominal pain, blood or mucus in stool with or without fever) and of bowel perforation (ie, peritoneal signs and ileus).</li> <li>Participants with ≥ Grade 2 diarrhea</li> </ul> | |
| | Grade 4 | Permanently discontinue | | <ul> <li>suspecting colitis should consider GI consultation and performing endoscopy to rule out colitis.</li> <li>Participants with diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion.</li> </ul> | |

Product: MK-3475 31 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

#### **General Instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤10 mg prednisone or equivalent per day within 12 weeks.
- **3.** For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with corticosteroid and/or other therapies | Monitor and follow-up |
|---|---|---|---|---|
| AST / ALT<br>elevation or<br>Increased | Grade 2 | Withhold | Administer corticosteroids (initial<br>dose of 0.5- 1 mg/kg prednisone or<br>equivalent) followed by taper | Monitor with liver function tests (consider<br>weekly or more frequently until liver<br>enzyme value returned to baseline or is |
| bilirubin | Grade 3 or 4 | Permanently discontinue | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | stable |
| Type 1 diabetes<br>mellitus (T1DM)<br>or<br>Hyperglycemia | Newly onset T1DM or Grade 3 or 4 hyperglycemia associated with evidence of β-cell failure | Withhold | <ul> <li>Initiate insulin replacement therapy for participants with T1DM</li> <li>Administer anti-hyperglycemic in participants with hyperglycemia</li> </ul> | Monitor participants for hyperglycemia or<br>other signs and symptoms of diabetes. |
| Hypophysitis | Grade 2 | Withhold | Administer corticosteroids and<br>initiate hormonal replacements as<br>clinically indicated. | Monitor for signs and symptoms of<br>hypophysitis (including hypopituitarism and<br>adrenal insufficiency) |
| | Grade 3 or 4 | Withhold or permanently discontinue <sup>1</sup> | , | |
| Hyperthyroidism | Grade 2 | Continue | | Monitor for signs and symptoms of thyroid disorders. |

Product: MK-3475
27Jan2022

#### **General Instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤10 mg prednisone or equivalent per day within 12 weeks.
- 3. For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with corticosteroid and/or other therapies | Monitor and follow-up |
|---|---|---|---|---|
| | Grade 3 or 4 | Withhold or permanently discontinue <sup>1</sup> | Treat with non-selective beta-<br>blockers (eg, propranolol) or<br>thionamides as appropriate | |
| Hypothyroidism | Grade 2-4 | Continue | Initiate thyroid replacement<br>hormones (eg, levothyroxine or<br>liothyroinine) per standard of care | Monitor for signs and symptoms of thyroid disorders. |
| Nephritis and<br>Renal | Grade 2 | | Monitor changes of renal function | |
| dysfunction | Grade 3 or 4 | Permanently discontinue | equivalent) followed by taper. | |
| Myocarditis | Grade 1 or 2 | Withhold | Based on severity of AE administer corticosteroids | Ensure adequate evaluation to confirm<br>etiology and/or exclude other causes |
| | Grade 3 or 4 | Permanently discontinue | | |
| All other immune-related | Intolerable/<br>persistent Grade 2 | Withhold | Based on type and severity of AE administer corticosteroids | Ensure adequate evaluation to confirm etiology and/or exclude other causes |
| AEs | Grade 3 | Withhold or<br>discontinue based<br>on the type of<br>event. Events that<br>require<br>discontinuation | | |

Product: MK-3475
27Jan2022

#### **General Instructions:**

- 1. Corticosteroid taper should be initiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks.
- 2. For situations where pembrolizumab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and corticosteroid has been tapered. Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or corticosteroids cannot be reduced to ≤10 mg prednisone or equivalent per day within 12 weeks.
- 3. For severe and life-threatening irAEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment should be initiated if irAEs cannot be controlled by corticosteroids.

| Immune-related<br>AEs | Toxicity grade or conditions (CTCAEv4.0) | Action taken to pembrolizumab | irAE management with corticosteroid and/or other therapies | Monitor and follow-up |
|---|---|---|---|---|
| | Grade 4 or recurrent Grade 3 | include and not limited to: Gullain-Barre Syndrome, encephalitis Permanently discontinue | | |

1. Withhold or permanently discontinue pembrolizumab is at the discretion of the investigator or treating physician.

#### **NOTE:**

For participants with Grade 3 or 4 immune-related endocrinopathy where withhold of pembrolizumab is required, pembrolizumab may be resumed when AE resolves to  $\leq$  Grade 2 and is controlled with hormonal replacement therapy or achieved metabolic control (in case of T1DM).

Product: MK-3475


34

Dosing interruptions are permitted in the case of medical / surgical events or logistical reasons not related to study therapy (e.g., elective surgery, unrelated medical events, patient vacation, and/or holidays). Subjects should be placed back on study therapy within 3 weeks of the scheduled interruption, unless due to socio-economic reasons (e.g. insurance-related issues) and unless otherwise discussed with the IND Sponsor. The reason for interruption should be documented in the patient's study record.

## **5.2.2** Timing of Dose Administration

Trial treatment should be administered on Day 1 of each 21-day cycle after all procedures/assessments have been completed as detailed on the Trial Flow Chart (Section 6.0). Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

All trial treatments will be administered on an outpatient basis.

Pembrolizumab (MK-3475) 200 mg will be administered as a 30 minute IV infusion every 3 weeks (21 days). Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).

The Pharmacy Manual contains specific instructions for the preparation of the pembrolizumab infusion fluid and administration of infusion solution.

## 5.2.3 Continuing Study Drug Administration after Initial Evidence of Radiologic Disease Progression

Immunotherapeutic agents such as pembrolizumab (MK-3475) may produce antitumor effects by potentiating endogenous cancer-specific immune responses. The response patterns seen with such an approach may extend beyond the typical time course of responses seen with cytotoxic agents, and can manifest as a clinical response after an initial increase in tumor burden or even the appearance of new lesions.

If initial radiologic imaging shows PD, tumor assessment should be repeated ≥4 weeks later in order to confirm PD with the option of continuing treatment per below while awaiting radiologic confirmation of progression. If repeat imaging shows a reduction in the tumor burden compared to the initial scan demonstrating PD, treatment may be continued as per treatment calendar. If repeat imaging confirms progressive disease, subjects will be discontinued from study therapy (exception noted in Section 7.1.2.5.1). In determining whether or not the tumor burden has increased or decreased, Investigators should consider all target lesions as well as non-target lesions (please refer to the Procedures Manual).

When feasible, subjects should not be discontinued until progression is confirmed; however,

Product: MK-3475

Product: MK-3475
27Jan2022

the decision to continue study treatment after the 1st evidence of disease progression is at the Investigator's discretion based on the clinical status of the subject as described in Table 4 below. Subjects may receive study treatment while waiting for confirmation of PD if they are clinically stable as defined by the following criteria:

- Absence of signs and symptoms (including worsening of laboratory values) indicating disease progression
- No decline in ECOG performance status
- Absence of rapid progression of disease
- Absence of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention.

Table 4 Imaging and Treatment After 1st Radiologic Evidence of PD

| | Clinically Stable | | Clinically Unstable | |
|---|---|---|---|---|
| | Imaging | Treatment | Imaging | Treatment |
| 1 <sup>st</sup> radiologic<br>evidence of PD | Repeat imaging<br>at ≥4 weeks to<br>confirm PD | May continue<br>study treatment at<br>the Investigator's<br>discretion while<br>awaiting<br>confirmatory scan | Repeat imaging at ≥4 weeks to confirm PD if possible | Discontinue treatment |
| Repeat scan confirms PD | No additional imaging required | Discontinue treatment (exception noted in Section 7.1.2.5) | No additional imaging required | N/A |
| Repeat scan<br>shows SD, PR<br>or CR | Continue<br>regularly<br>scheduled<br>imaging<br>assessments<br>every 9 weeks | Continue study<br>treatment at the<br>Investigator's<br>discretion | Continue<br>regularly<br>scheduled<br>imaging<br>assessments<br>every 9 weeks | May restart<br>study treatment<br>if condition has<br>improved and/or<br>clinically stable<br>per<br>Investigator's<br>discretion |

## 5.2.4 Trial Blinding/Masking

This is an open-label trial; therefore, the IND Sponsor, investigator and subject will know the treatment administered.

#### 5.3 Randomization or Treatment Allocation

Subjects participating in this trial will be allocated by non-random assignment.

Product: MK-3475

36 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

#### 5.4 Stratification

No stratification based on age, gender, or other characteristics will be used in this trial.

#### 5.5 **Concomitant Medications/Vaccinations (Allowed & Prohibited)**

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for one of these or other medications or vaccinations specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Merck Clinical team. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician.

Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

## **5.5.1** Acceptable Concomitant Medications

All treatments that the investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the electronic medical record (EMR) including all prescription, over-the-counter (OTC), and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date may also be included on the EMR.

All concomitant medications received within 28 days before the first dose of trial treatment and 30 days after the last dose of trial treatment should be recorded. Concomitant medications administered after 30 days after the last dose of trial treatment should be recorded if associated with SAEs and ECIs as defined in Section 7.2.

#### **5.5.2** Prohibited Concomitant Medications

Subjects are prohibited from receiving the following therapies during the Screening and Treatment Phase (including retreatment for post-complete response relapse) of this trial:

- Antineoplastic systemic chemotherapy or biological therapy
- Immunotherapy not specified in this protocol
- Chemotherapy not specified in this protocol
- Investigational agents other than pembrolizumab
- Radiation therapy
  - o Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be allowed at the investigator's discretion.
Product: MK-3475 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.

37

- Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the IND Sponsor.
- Herbal products.

Subjects who, in the assessment by the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the trial. Subjects may receive other medications that the investigator deems to be medically necessary.

The Exclusion Criteria describes other medications which are prohibited in this trial.

There are no prohibited therapies during the Post-Treatment Follow-up Phase.

#### **Rescue Medications & Supportive Care** 5.6

### **5.6.1 Supportive Care Guidelines**

Subjects should receive appropriate supportive care measures as deemed necessary by the treating investigator. Suggested supportive care measures for the management of adverse events with potential immunologic etiology are outlined below. Where appropriate, these guidelines include the use of oral or intravenous treatment with corticosteroids as well as additional anti-inflammatory agents if symptoms do not improve with administration of corticosteroids. Note that several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased. For each disorder, attempts should be made to rule out other causes such as metastatic disease or bacterial or viral infection, which might require additional supportive care. The treatment guidelines are intended to be applied when the investigator determines the events to be related to pembrolizumab.

Note: if after the evaluation the event is determined not to be related, the investigator does not need to follow the treatment guidance (as outlined below). Refer to Section 5.2.1 for dose modification.

It may be necessary to perform conditional procedures such as bronchoscopy, endoscopy, or skin photography as part of evaluation of the event.

#### **Pneumonitis:**

o For Grade 2 events, treat with systemic corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

Product: MK-3475


27Jan2022

• For **Grade 3-4 events**, immediately treat with intravenous steroids. Administer additional anti-inflammatory measures, as needed.

o Add prophylactic antibiotics for opportunistic infections in the case of prolonged steroid administration.

### Diarrhea/Colitis:

Subjects should be carefully monitored for signs and symptoms of enterocolitis (such as diarrhea, abdominal pain, blood or mucus in stool, with or without fever) and of bowel perforation (such as peritoneal signs and ileus).

- O All subjects who experience diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion. For Grade 2 or higher diarrhea, consider GI consultation and endoscopy to confirm or rule out colitis.
- o For **Grade 2 diarrhea/colitis** that persists greater than 3 days, administer oral corticosteroids.
- For **Grade 3 or 4 diarrhea/colitis** that persists > 1 week, treat with intravenous steroids followed by high dose oral steroids.
- O When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

# • Type 1 diabetes mellitus (if new onset, including diabetic ketoacidosis [DKA]) or ≥ Grade 3 Hyperglycemia, if associated with ketosis (ketonuria) or metabolic acidosis (DKA)

- o For **T1DM** or **Grade 3-4** Hyperglycemia
  - Insulin replacement therapy is recommended for Type I diabetes mellitus and for Grade 3-4 hyperglycemia associated with metabolic acidosis or ketonuria.
  - Evaluate patients with serum glucose and a metabolic panel, urine ketones, glycosylated hemoglobin, and C-peptide.

### • Hypophysitis:

- o For **Grade 2** events, treat with corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.
- o For **Grade 3-4** events, treat with an initial dose of IV corticosteroids followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

# • Hyperthyroidism or Hypothyroidism:

Thyroid disorders can occur at any time during treatment. Monitor patients for changes in thyroid function (at the start of treatment, periodically during treatment, and as indicated based on clinical evaluation) and for clinical signs and symptoms of thyroid disorders.


**Grade 2** hyperthyroidism events (and **Grade 2-4** hypothyroidism):

- In hyperthyroidism, non-selective beta-blockers (e.g. propranolol) are suggested as initial therapy.
- In hypothyroidism, thyroid hormone replacement therapy, with levothyroxine or liothyroinine, is indicated per standard of care.
- **Grade 3-4** hyperthyroidism
  - Treat with an initial dose of IV corticosteroid followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

### Hepatic:

- For Grade 2 events, monitor liver function tests more frequently until returned to baseline values (consider weekly).
  - Treat with IV or oral corticosteroids
- o For **Grade 3-4** events, treat with intravenous corticosteroids for 24 to 48 hours.
- When symptoms improve to Grade 1 or less, a steroid taper should be started and continued over no less than 4 weeks.

### **Renal Failure or Nephritis:**

- o For Grade 2 events, treat with corticosteroids.
- o For **Grade 3-4** events, treat with systemic corticosteroids.
- o When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

Management of Infusion Reactions: Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion.

Table 5 below shows treatment guidelines for subjects who experience an infusion reaction associated with administration of pembrolizumab (MK-3475).

Table 5 Infusion Reaction Treatment Guidelines

| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |
| Grade 2 | Stop Infusion and monitor symptoms. | Subject may be premedicated 1.5h |
| Requires infusion interruption but | Additional appropriate medical therapy may | (± 30 minutes) prior to infusion of |
| responds promptly to symptomatic | include but is not limited to: | pembrolizumab (MK-3475) with: |
| treatment (e.g., antihistamines, | IV fluids | |
| NSAIDS, narcotics, IV fluids); | Antihistamines | Diphenhydramine 50 mg po (or |
| prophylactic medications indicated for | NSAIDS | equivalent dose of antihistamine). |
| <=24 hrs | Acetaminophen | |
| | Narcotics | Acetaminophen 500-1000 mg po |
| | | (or equivalent dose of antipyretic). |

Product: MK-3475 40 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. If symptoms resolve within one hour of stopping drug infusion, the infusion may be restarted at 50% of the original infusion rate (e.g., from 100 mL/hr to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and the subject should be premedicated for the next scheduled dose. Subjects who develop Grade 2 toxicity despite adequate premedication should be permanently discontinued from further trial | |
| | treatment administration. | |
| Grades 3 or 4 Grade 3: Prolonged (i.e., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for other clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Stop Infusion. Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines NSAIDS Acetaminophen Narcotics Oxygen Pressors Corticosteroids Epinephrine | No subsequent dosing |
| Grade 4:<br>Life-threatening; pressor or ventilatory<br>support indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. Hospitalization may be indicated. Subject is permanently discontinued from further trial treatment administration. | |

# 5.7 Diet/Activity/Other Considerations

### 5.7.1 Diet

Subjects should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea or vomiting.

### 5.7.2 Contraception

Pembrolizumab may have adverse effects on a fetus in utero. Furthermore, it is not known if pembrolizumab has transient adverse effects on the composition of sperm. Non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive. Highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is ≥45 years of age and has not had menses for greater than 1 year will be considered postmenopausal), or 3) not heterosexually active for the duration of the study. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should

Product: MK-3475


41

start using birth control from study Visit 1 throughout the study period up to 120 days after the last dose of study therapy.

The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

Subjects should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study. In order to participate in the study they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period defined in <a href="Section 7.2.2">Section 7.2.2</a>-Reporting of Pregnancy and Lactation to the IND Sponsor and to Merck. If there is any question that a subject will not reliably comply with the requirements for contraception, that subject should not be entered into the study.

### 5.7.3 Use in Pregnancy

If a subject inadvertently becomes pregnant while on treatment with pembrolizumab, the subject will immediately be removed from the study. The site will contact the subject at least monthly and document the subject's status until the pregnancy has been completed or terminated. The outcome of the pregnancy will be reported to the IND Sponsor and to Merck without delay and within 24 hours to the IND Sponsor and within 2 working days to Merck if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn).

The study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn to the IND Sponsor. If a male subject impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported to the IND Sponsor and to Merck and followed as described above and in Section 7.2.2.

### 5.7.4 Use in Nursing Women

It is unknown whether pembrolizumab is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, subjects who are breast-feeding are not eligible for enrollment.

### 5.8 Subject Withdrawal/Discontinuation Criteria

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the discretion of the investigator should any untoward effect occur. In addition, a subject may be withdrawn by the investigator if enrollment into the trial is inappropriate, the trial plan is

Product: MK-3475


violated, or for administrative and/or other safety reasons. Specific details regarding discontinuation or withdrawal are provided in Section 7.1.4 – Other Procedures. Subjects who have attained a confirmed CR that have been treated for at least 27 weeks (9 cycles) with pembrolizumab and had at least two treatments with pembrolizumab beyond the date when the initial CR was declared may also consider discontinuation of treatment, details for which are provided in Section 5.8.1.

A subject must be discontinued from the trial for any of the following reasons:

- The subject or legal representative (such as a parent or legal guardian) withdraws consent.
- Confirmed radiographic disease progression

*Note*: For unconfirmed radiographic disease progression, please see <u>Section 7.1.2.5</u>.

*Note*: A subject may be granted an exception to continue on treatment with confirmed radiographic progression if clinically stable or clinically improved, please see Section 7.1.2.5.

- Clinical progression as determined by PI or treating physician.
- Unacceptable adverse experiences as described in <u>Section 5.2.1.2</u>
- Intercurrent illness that prevents further administration of treatment
- Investigator's decision to withdraw the subject
- The subject has a confirmed positive serum pregnancy test
- Noncompliance with trial treatment or procedure requirements
- The subject is lost to follow-up
- Completed 24 months of uninterrupted treatment with pembrolizumab or 34 administrations of study medication, whichever is later. A patient may continue past 24 months (or 34 administrations) after discussion with Merck on a case by case basis.

Note: 24 months of study medication is calculated from the date of first dose. Subjects who stop pembrolizumab after 24 months may be eligible for up to one year of additional study treatment if they progress after stopping study treatment provided they meet the requirements detailed in Section 7.1.5.5

• Administrative reasons

Product: MK-3475

43 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

The End of Treatment and Follow-up visit procedures are listed in <u>Section 6</u> (Protocol Flow Chart) and Section 7.1.5 (Visit Requirements). After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment as described in Section 7.2.3.1). Subjects who discontinue for reasons other than progressive disease will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent or becoming lost to follow-up. After documented disease progression each subject will be followed by telephone or chart review for overall survival until death, withdrawal of consent, or the end of the study, whichever occurs first.

#### Discontinuation of Study Therapy after CR 5.8.1

Discontinuation of treatment may be considered for subjects who have attained a confirmed CR that have been treated for at least 27 weeks (9 cycles) with pembrolizumab and had at least two treatments with pembrolizumab beyond the date when the initial CR was declared. Subjects who then experience radiographic disease progression may be eligible for up to one year of additional treatment with pembrolizumab via the Second Course Phase at the discretion of the investigator if no cancer treatment was administered since the last dose of pembrolizumab, the subject meets the safety parameters listed in the Inclusion/Exclusion criteria, and the trial is open. Subjects will resume therapy at the same dose and schedule at the time of initial discontinuation. Additional details are provided in Section 7.1.5.5.

#### 5.9 **Subject Replacement Strategy**

Patients will not be replaced on study. However, if a patient is considered to be non-evaluable for primary efficacy assessment (alive and progression free at 27 weeks), additional subjects may be enrolled in a given cohort to ensure that the required number of evaluable subjects in each cohort is achieved.

### 5.10 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

- 1. Quality or quantity of data recording is inaccurate or incomplete
- 2. Poor adherence to protocol and regulatory requirements
- 3. Incidence or severity of adverse drug reaction in a particular cohort or other studies indicates a potential health hazard to subjects
- 4. Plans to modify or discontinue the development of the study drug

In the event of Merck decision to no longer supply study drug, ample notification will be provided so that appropriate adjustments to subject treatment can be made.

Product: MK-3475 44

# 6.0 TRIAL FLOW CHART

# 6.1 Study Flow Chart

| Trial Period: | Screening<br>Phase | | | Tr | eatmen | t Cycle | es <sup>a</sup> | | | End of<br>Treatment | | Post-Treatme | ent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Screening | 1 | 2 | 3 | 4 | To b | | ited bey<br>8 cycle | | Discon | Safety<br>Follow- | Follow-up | Survival |
| Cycle/Title: | (Visit 1) | | | | | 5 | 6 | 7 | 8 | | up | Visits <sup>c</sup> | Follow-up |
| Scheduling Window<br>(Days): | -28 to -1 | Day 1<br>(-3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | At time<br>of<br>Discon | 30 days<br>from<br>last<br>dose<br>(± 7 days) | Post<br>discon<br>(± 7 days) | Every<br>12<br>weeks<br>(± 4 weeks) |
| Administrative Procedures | | | | | | | | | | | | | |
| Informed Consent <sup>b</sup> | $X^b$ | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | | | | | | | |
| Demographics and Medical History | X | | | | | | | | | | | | |
| Concomitant Medication Review | X <sup>d</sup> | X | X | X | X | X | X | X | X | X | $X^d$ | X | |
| Trial Treatment Administration <sup>a</sup> | | X | X | X | X | X | X | X | X | | | | |
| Post-study Anticancer Therapy Status | | | | | | | | | | | | X | X |
| Survival Status | | | | | | | | | | | | | X <sup>X</sup> |
| Clinical Procedures/Assessments | | | | | | | | 3 | - | | | • | |
| Review Adverse Events <sup>e</sup> | X | X | X | X | X | X | X | X | X | X | Xe | Xe | |
| Physical Examination <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| Vital Signs and Weight <sup>g</sup> | X | Xg | X | X | X | X | X | X | X | X | X | X | |
| ECOG Performance Status | X | X | X | X | X | X | $X^h$ | Xh | Xh | X | X | X | |
| Laboratory Procedures/Assessments: analysis per | formed by LO | CAL la | borato | ry | | | | | | | | | |
| Pregnancy Test – Urine or Serum β-HCG <sup>i</sup> | Xi | X | X | X | X | X | X | X | X | X | | | |
| PT/INR and aPTT | $\mathbf{X}^{\mathrm{j}}$ | | As Clinically Indicated | | | | | | | | | | |
| CBC with Differentialk | $\mathbf{X}^{\mathrm{j}}$ | $X^k$ | X | X | X | X | X | X | X | X | X <sup>n</sup> | X | |

Product: MK-3475 45 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

| Trial Period: | Screening<br>Phase | | | Tr | eatmen | t Cycle | es <sup>a</sup> | | | End of<br>Treatment | ] | Post-Treatme | nt |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Screening | 1 | 1 2 3 | | 4 | To be repeated beyond 8 cycles <sup>a</sup> | | | | Discon | Safety<br>Follow- | Follow-up | Survival |
| Cycle/Title: | (Visit 1) | | | | | 5 | 6 | 7 | 8 | | up | Visits <sup>c</sup> | Follow-up |
| Scheduling Window (Days): | -28 to -1 | Day 1<br>(-3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | At time<br>of<br>Discon | 30 days<br>from<br>last<br>dose<br>(± 7 days) | Post<br>discon<br>(± 7 days) | Every<br>12<br>weeks<br>(± 4 weeks) |
| Comprehensive Chemistry Panel <sup>k</sup> | $\mathbf{X}^{\mathrm{j}}$ | $X^k$ | X | X | X | X | X | X | X | X | X <sup>n</sup> | X | |
| Urinalysis <sup>k,l</sup> | $\mathbf{X}^{\mathrm{j}}$ | | | | $X^{l}$ | | | $X^{l}$ | | | X <sup>n</sup> | | |
| T3, FT4 and TSH <sup>k</sup> | $\mathbf{X}^{\mathrm{j}}$ | | | | $X^{l}$ | | | $X^{l}$ | | | X <sup>n</sup> | | |
| Tumor Marker Assessment (if available) m | Хј | | | | Xm | | | Xm | | X <sup>m</sup> | | X <sup>m</sup> | |
| Efficacy Measurements | | | | | | | | | | | | | |
| Tumor Imaging <sup>a,o, p, q</sup> | X <sup>W</sup> | | | | X | | | X | | $X^q$ | | X <sup>c</sup> | |
| Correlative Studies | | | | | | | | | | | | | |
| Tissue Collection for PD-L1 Characterization <sup>r</sup> | X <sup>r</sup> | | | | | | | | | | | | |
| Tumor Biopsy Tissue Collection | Xs | Xs | | | | | | | | Xs | | | |
| PBMC Collection <sup>t</sup> | X | X <sup>t</sup> | | | X | | | X | | X <sup>t</sup> | | | |
| Immune-related Imaging | X <sup>u</sup> | | | | Xu | | | Xu | | X <sup>u</sup> | | | |
| Patient-Reported Outcomes | | | | 1 | • | | | | | | | | |
| PRO-CTCAE Questionnaires <sup>v</sup> | X | Weekl | y for 9 | Weeks | Weeks Every 2 Weeks until Week 54, then every 4 Weeks | | | X | | | | | |

a. Treatment cycles are 3 weeks (21 days). Radiographic imaging should be performed every 9 weeks (3 cycles or 63 days ± 7 days) regardless of any treatment delays (i.e. Screening visit, after to Cycle 3, Cycle 6, Cycle 9 and then every 3 cycles (9 weeks)). However, after 6 months, at the physician's discretion, if patients have had CR, PR or SD > 27 weeks, then radiographic imaging may be performed every 12 weeks (4 cycles or 84 days ± 7 days).

b. Written consent must be obtained prior to performing any protocol specific procedure. Results of a test performed prior to the subject signing consent as part of routine clinical management are acceptable in lieu of a screening test if performed within the specified time frame (e.g., within 28 days prior to the first dose of trial treatment). Baseline number will be assigned when the study informed consent is signed.

c. The Follow-Up Visits post discontinuation may be performed every 9 weeks, 12 weeks, or at the discretion of the treating physician. In subjects who discontinue study

Product: MK-3475 46 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

| Trial Period: | Screening<br>Phase | | Treatment Cycles <sup>a</sup> | | | | | End of<br>Treatment | ] | Post-Treatment | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | | 1 | 1 2 | | 1 2 | | 1 2 | | 1 2 | 1 2 | 2 | 2 3 | 4 | To be repeated beyond 8 cycles <sup>a</sup> | Discon | Safety<br>Follow- | Follow-up | Survival |
| Cycle/Title: | (Visit 1) | | | - | | 5 | 6 | 7 | 8 | | up | Visits <sup>c</sup> | Follow-up | | | | | |
| Scheduling Window (Days): | | Day 1<br>(-3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | 1<br>(± 3 | of<br>Discon | 30 days<br>from<br>last<br>dose<br>(± 7 days) | Post<br>discon<br>(± 7 days) | Every<br>12<br>weeks<br>(± 4 weeks) | | | | | |

therapy without documented disease progression, every effort should be made to continue monitoring their disease status by radiologic imaging every 9 weeks (± 7 days) until (1) the start of new anti-cancer treatment, (2) documented radiological or clinical disease progression, (3) death, or (4) the end of the study, whichever occurs first.

- d. Prior medications Record all medications taken 28 days before the first dose of trial treatment. Concomitant medications Enter new medications started during the trial and 30 days after last dose of trial treatment regardless of when the Safety Follow-up visit occurs.
- e. Patients enrolled on this study will be approached for co-enrollment on PA15-0315 prospective study to assess immune-related adverse events when receiving immunotherapy All samples and scans will be collected using procedures characterized in this protocol and all patients will be consented for procedures done under this optional protocol separately. Record all AEs occurring within 30 days after the last dose of trial treatment regardless of when the Safety Follow-up visit occurs. After 30 days, record all SAEs (related and unrelated to trial treatment) / ECIs occurring up to 90 days after the last dose of trial treatment or the start of new anti-cancer treatment, whichever comes first. Afterwards, any drug related AE regardless of seriousness occurring outside of any reporting timeframes must be reported
- f. Physical exams are to be completed at screening, Day 1 of every Cycle, End of Treatment, Safety Follow-up and every 9 week Follow-up visits.
- g. Height will be measured at visit 1 only.
- h. Following Cycle 8, the ECOG performance status should be determined only in conjunction with a protocol-specified full or directed physical exam (Cycle 9, 11, 13, 15, 17, 19 and every 2 cycles thereafter.
- i. For women of reproductive potential, a urine pregnancy test should be performed within 72 hours prior to first dose of trial treatment. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test performed by the local study site laboratory will be required. Pregnancy tests (serum and/or urine tests) should be repeated if required by local guidelines.
- Laboratory tests for screening are to be performed within 28 days prior to the first dose of trial treatment.
- k. After Cycle 1, lab samples can be collected up to 72 hours (3 days) prior to the scheduled time point.
- 1. Urinalysis and T3, FT4 and TSH are to be repeated every 3 cycles at the time of restaging. If the urinalysis is abnormal, a microscopic urinalysis will be performed.
- m. Tumor marker assessment is not an additional study-related laboratory evaluation. The purpose is to collect information that may be a part of standard clinical assessment for certain tumor types. Data collection (if applicable and if available) should occur every 9 weeks (3 cycles or 63 days ± 7 days) regardless of any treatment delays (i.e. Screening visit, after to Cycle 3, Cycle 6, Cycle 9 and then every 3 or 4 cycles (9 or 12 weeks) thereafter coinciding with imaging visits). Upon discontinuation, tumor marker data collection will occur every 9 or 12 weeks coinciding with post-treatment imaging follow-up visits.
- n. Unresolved abnormal labs that are drug related AEs should be followed until resolution.
- o. The initial tumor imaging will be performed within 28 days prior to the first dose of trial treatment. Scans performed as part of routine clinical management are acceptable for use as the screening scan if they are of diagnostic quality and performed within 28 days prior to the first dose of trial treatment. On-study imaging will be performed every 9 weeks (± 7 days) after the first dose of trial treatment and should follow calendar days and should not be adjusted for delays in cycle starts or withholding of pembrolizumab (MK-3475) cycle frequencies. However, after 6 months, at the physician's discretion, if patients have had CR, PR or SD > 27 weeks, then radiographic imaging may be performed every 12 weeks (4 cycles or 84 days ± 7 days). The same imaging technique should be used in a subject throughout the trial. Local reading (investigator assessment

Product: MK-3475
27Jan2022

| Trial Period: | Screening<br>Phase | Treatment Cycles <sup>a</sup> | | | | | End of<br>Treatment | Post-Treatment | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | U | | | | 4 | Tol | o be repeated beyond<br>8 cycles <sup>a</sup> | | | Discon | HOLLOW | Follow-up | 1 |
| Cycle/Title: | (Visit 1) | | | | | 5 | 6 | 7 | 8 | | up | Visits <sup>c</sup> | Follow-up |
| Scheduling Window<br>(Days): | | Day 1<br>(-3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days) | Day<br>1<br>(± 3<br>days | Day<br>1<br>(± 3<br>days) | 1<br>(± 3 | 1<br>(± 3 | of<br>Discon | 30 days<br>from<br>last<br>dose<br>(± 7 days) | Post<br>discon<br>(± 7 days) | Every<br>12<br>weeks<br>(± 4 weeks) |

with site radiology reading) will be used to determine eligibility and for subject management. Tumor imaging and assessment per local standard of care should be performed for patient management, and may include additional imaging (e.g. bone scan for prostate cancer patients) and appropriate tumor markers.

- p. Per the modified RECIST 1.1 or irRECIST used in this protocol, if imaging shows progressive disease, the imaging assessment should be repeated at a minimum of 4 weeks later in order to confirm progressive disease.
- q. If a scan was obtained within 4 weeks prior to the date of discontinuation, then a scan at treatment discontinuation isn't mandatory. In subjects who discontinue study therapy without confirmed disease progression, a radiological evaluation should be repeated at the time of treatment discontinuation (i.e. date of discontinuation ± 4 week window).
- r. Mandatory archived or newly obtained (within 42 days (6 weeks)) FFPE (formalin-fixed paraffin embedded) for 5 unstained (4 or 5 micron, 4 micron preferred) slides must be submitted for characterization at a central lab for PD-L1 characterization. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Tumor lesions not previously irradiated must be provided (tumors progressing in a prior site of radiation are allowed for PD-L1 characterization).
- s. Tumor tissue will be obtained pre- treatment (baseline), between Cycle 1 Day 15 and Cycle 1 Day 21, and at progression (if patient had CR, PR or SD > 27 weeks) provided there is technically biopsiable tumor, and it is safe for patient to undergo biopsy. In Cohort 9: Paraganglioma-pheochromocytoma or Cohort 10, where there is prominent bony disease, biopsies may not be possible due to the nature of the disease.
- t. Peripheral blood mononuclear cell (PBMC) will be collected at baseline, tumor restaging, in conjunction with biopsies, and time of progression (if patients have had CR/PR/or SD for > 27 weeks). PBMC collections at tumor restaging and in conjunction with biopsies will have a +/- 1 day window.
- u. The CT or MRI tumor scans for tumor assessment will be utilized for immune-related imaging correlatives. Additional scans will not be required.
- v. Baseline questionnaires will be performed in person with the study team. Subsequent questionnaires will be issued weekly for 9 weeks and every 2 week until Week 54, and every 4 weeks thereafter until the End of Treatment or up to Week 81. All questionnaires will have a +/-2 day window.
- w. Subjects in Cohort 2 (small cell malignancies of non-pulmonary origin) are required to have confirmation of no brain metastases via imaging at screening.
- x. Investigators will collect survival data for patients after progression of disease unless patient fully withdrew consent to participate in the study using information from a chart review, patient visit, or telephone call.

Product: MK-3475


48

### 7.0 TRIAL PROCEDURES

#### 7.1 Trial Procedures

The Trial Flow Chart - Section 6.0 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below. It may be necessary to perform these procedures at unscheduled time points if deemed clinically necessary by the investigator.

Furthermore, additional evaluations/testing may be deemed necessary by the IND Sponsor and/or Merck for reasons related to subject safety. In some cases, such evaluation/testing may be potentially sensitive in nature (e.g., HIV, Hepatitis C, etc.), and thus local regulations may require that additional informed consent be obtained from the subject. In these cases, such evaluations/testing will be performed in accordance with those regulations.

#### 7.1.1 Administrative Procedures

#### 7.1.1.1 Informed Consent

The Investigator must obtain documented consent from each potential subject prior to participating in a clinical trial.

#### 7.1.1.1 General Informed Consent

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the subject before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB/ERC requirements, applicable laws and regulations and IND Sponsor requirements.

Product: MK-3475


49

For patients enrolled on this study prior to approval of Protocol Version 13, the baseline blood samples collected for correlative research studies may be used for the germline DNA testing under the Waiver of Consent. All patients consent to the blood collection for the correlative blood testing. Patients off-study prior to Version 13 would not be able to be reconsented. The purpose of Protocol Version 13 was to specify an additional type of testing. Under the Waiver of Consent, samples from patients no longer on the study will be used for the specific germline DNA testing. Samples from patients that withdrew consent will not be used.

For patients enrolled on this study prior to approval of Protocol Version 14 that cannot be reconsented, survival data, de-identified clinical data and RNA sequencing data output, imaging, and baseline plasma samples collected for translational research studies may be used under the Waiver of Consent for entities listed in the 10.1.4 Data Sharing section of the protocol. All patients consented to the collection of data and blood for translational research. Patients off-study prior to Version 14 would not be able to be reconsented. Under the Waiver of Consent, samples from patients no longer on the study will be used for testing conducted by entities listed in 10.1.4 Data Sharing. Samples and data from patients that withdrew consent will not be used for these purposes.

### 7.1.1.2 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the trial.

### 7.1.1.3 Medical History

A medical history will be obtained by the investigator or qualified designee. Medical history will include all active conditions, and any condition diagnosed within the prior 10 years that are considered to be clinically significant by the Investigator. Details regarding the disease for which the subject has enrolled in this study will be recorded separately and not listed as medical history.

#### 7.1.1.4 Prior and Concomitant Medications Review

### 7.1.1.4.1 Prior Medications

The investigator or qualified designee will review prior medication use, including any protocol-specified washout requirement, and record prior medication taken by the subject within 28 days before starting the trial. Treatment for the disease for which the subject has enrolled in this study will be recorded separately and not listed as a prior medication.

Product: MK-3475

Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

50

### 7.1.1.4.2 Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the subject during the trial. All medications related to reportable SAEs and ECIs should be recorded as defined in Section 7.2.

#### 7.1.1.5 Disease Details and Treatments

#### 7.1.1.5.1 Disease Details

The investigator or qualified designee will obtain prior and current details regarding disease status.

### 7.1.1.5.2 Prior Treatment Details

The investigator or qualified designee will review all prior cancer treatments including systemic treatments, radiation and surgeries.

### 7.1.1.5.3 Subsequent Anti-Cancer Therapy Status

The investigator or qualified designee will review all new anti-neoplastic therapy initiated after the last dose of trial treatment. If a subject initiates a new anti-cancer therapy within 30 days after the last dose of trial treatment, the 30 day Safety Follow-up visit must occur before the first dose of the new therapy. Once new anti-cancer therapy has been initiated the subject will move into survival follow-up.

### 7.1.1.6 Assignment of Screening Number

Consented subjects will not be given a unique screening number for randomization or allocation. All patients who meet eligibility criteria and are enrolled in this trial will be registered in Clinical Oncology Research Database (CORe) at the University of Texas MD Anderson Cancer Center at Houston. Each patient will have a CORe accession number.

### 7.1.1.7 Assignment of Randomization Number

Subjects participating in this trial will be allocated by non-random assignment; therefore, a randomization number will not be assigned to patients.

### 7.1.1.8 Trial Compliance (Medication/Diet/Activity/Other)

Interruptions from the protocol specified treatment plan for greater than 12 weeks between pembrolizumab (MK-3475) doses due to toxicity require consultation between the investigator and the IND Sponsor and written documentation of the collaborative decision on subject management.

Product: MK-3475


51

Administration of trial medication will be witnessed by the investigator and/or trial staff. The total volume of trial treatment infused will be compared to the total volume prepared to determine compliance with each dose administered.

The instructions for preparing and administering pembrolizumab (MK-3475) will be provided in the Pharmacy Manual.

### 7.1.2 Clinical Procedures/Assessments

### 7.1.2.1 Adverse Event (AE) Monitoring

The investigator or qualified designee will assess each subject to evaluate for potential new or worsening AEs as specified in the Trial Flow Chart and more frequently if clinically indicated. Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 4.03 (see Section 11.2). Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

For subjects receiving treatment with pembrolizumab all AEs of unknown etiology associated with pembrolizumab exposure should be evaluated to determine if it is possibly an event of clinical interest (ECI) of a potentially immunologic etiology (termed immune-related adverse events, or irAEs).

Please refer to <u>Section 7.2</u> for detailed information regarding the assessment and recording of AEs.

### 7.1.2.2 Physical Exam

The investigator or qualified designee will perform a complete physical exam during the screening period. Clinically significant abnormal findings should be recorded as medical history. A physical exam should be performed during screening, Day 1 of every Cycle, End of Treatment, Safety Follow-Up, and every 9-week Follow-up Visit. After the first dose of trial treatment, new clinically significant abnormal findings should be recorded as AEs.

# 7.1.2.3 Vital Signs

The investigator or qualified designee will take vital signs at screening, prior to the administration of each dose of trial treatment and at treatment discontinuation as specified in the Trial Flow Chart (Section 6.0). Vital signs should include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.

Product: MK-3475

52 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

### 7.1.2.4 Eastern Cooperative Oncology Group (ECOG) Performance Scale

The investigator or qualified designee will assess ECOG status (Section 11.1) at screening, prior to the administration of each dose of trial treatment and discontinuation of trial treatment as specified in the Trial Flow Chart.

### 7.1.2.5 Tumor Imaging and Assessment of Disease

RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated will be applied by the site as the primary measure for assessment of tumor response and as a basis for all protocol guidelines related to disease status (e.g., discontinuation of study therapy).

RECIST v1.1 or irRECIST will be adapted as follows to account for the unique tumor response seen in this class of therapeutics. If imaging shows PD, tumor assessment should be repeated  $\geq 4$  weeks later in order to confirm PD with the option of continuing treatment for clinically stable subjects as discussed below in Table 6. Clinically stable is defined by the following criteria:

- Absence of signs and symptoms indicating disease progression
- No decline in ECOG performance status
- Absence of rapid progression of disease
- Absence of progressive tumor at critical anatomical sites (e.g., cord compression) requiring urgent alternative medical intervention.

Table 6 Imaging and Treatment after 1st Radiologic Evidence of PD

| | Clinical | ly Stable | Clinically | Unstable |
|---|---|---|---|---|
| | Imaging | Treatment | Imaging | Treatment |
| 1 <sup>st</sup> radiologic | Repeat imaging | May continue | Repeat imaging | Discontinue |
| evidence of PD | at $\geq$ 4 weeks to | study treatment | at $\geq$ 4 weeks to | treatment |
| | confirm PD | at the | confirm PD if | |
| | | Investigator's | possible | |
| | | discretion while | | |
| | | awaiting | | |
| | | confirmatory | | |
| | | scan | | |
| Repeat scan | No additional | Discontinue | No additional | N/A |
| confirms PD | imaging required | treatment | imaging required | |
| | | (exception noted | | |
| | | in <u>Section</u> | | |
| | | <u>7.1.2.5</u> .) | | |

27.Jan2022

Product: MK-3475

| Repeat scan | Continue | Continue study | Continue | May restart study |
|---|---|---|---|---|
| shows SD, PR | regularly | treatment at the | regularly | treatment if |
| or CR | scheduled | Investigator's | scheduled | condition has |
| | imaging | discretion | imaging | improved and/or |
| | assessments | | assessments | clinically stable |
| | every 9 weeks | | every 9 weeks | per Investigator's |
| | | | | discretion |

In determining whether or not the tumor burden has increased or decreased, Investigators should consider all target lesions as well as non-target lesions (please refer to the Procedures Manual). Subjects that are deemed clinically unstable are not required to have repeat imaging for confirmation. If radiologic progression is confirmed, then the subject will be discontinued from trial treatment. If radiologic progression is not confirmed, then the subject should resume/continue trial treatment and have their next scan according to the every 9 weeks  $(63 \text{ days} \pm 7 \text{ days})$ .

**NOTE**: If a subject with confirmed radiographic progression (i.e. 2 scans at least 28 days apart demonstrating progressive disease) is clinically stable or clinically improved, and there is no further increase in the tumor dimensions at the confirmatory scan, an exception may be considered to continue treatment upon consultation with the IND Sponsor. Clinically stable subjects should also have at the confirmatory scan no further increase in the target lesions, no unequivocal increase in non-target lesions, and no additional new lesions develop (non-worsening PD) to continue study treatment.

Local reading (investigator assessment with site radiology reading) based on RECIST v 1.1 or irRECIST will be used to determine subject eligibility and for subject management. Tumor imaging and assessment per local standard of care should be performed for patient management, and may include additional imaging (e.g. bone scan for prostate cancer patients) and appropriate tumor markers.

### 7.1.2.5.1 Initial Tumor Imaging

Initial tumor imaging must be performed within 28 days prior to the first dose of trial treatment. The site study team must review pre-trial images to confirm the subject has measurable disease per RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated. The baseline imaging scan should be submitted to the central imaging vendor for a possible retrospective analysis of this eligibility criterion.

Scans performed as part of routine clinical management are acceptable for use as the screening scan if they are of diagnostic quality and performed within 28 days prior to the first dose of trial treatment. The same imaging technique should be used in a subject throughout the study.

Product: MK-3475


54

### 7.1.2.5.2 Tumor Imaging During Trial

Tumor imaging may be performed by CT or magnetic resonance imaging (MRI), but the same imaging technique should be used in a subject throughout the trial. Imaging should be performed every 9 weeks (63 days  $\pm$  7 days) from the first dose of trial treatment or more frequently if clinically indicated. Imaging should not be delayed for delays in cycle starts or withholding of pembrolizumab (MK-3475) cycle intervals. After 6 months, at the physician's discretion, if patients have had CR, PR or SD > 27 weeks, then radiographic imaging may be performed every 12 weeks (4 cycles or 84 days  $\pm$  7 days).

Per RECIST 1.1 or irRECIST, response should be confirmed by a repeat radiographic assessment not less than 4 weeks from the date the response was first documented. The scan for confirmation of response may be performed at the earliest 4 weeks after the first indication of response, or at the next scheduled scan, whichever is clinically indicated.

Imaging should continue to be performed until documented disease progression, the start of new anti-cancer treatment, withdrawal of consent, death, or the end of the study, whichever occurs first. Disease progression should be confirmed at least 4 weeks after the first scan indicating progressive disease in clinically stable subjects. Subjects who have unconfirmed disease progression may continue on treatment until progression is confirmed provided they have met the conditions detailed in Section 7.1.2.5.

### 7.1.2.5.3 Tumor Imaging During Follow-Up

Imaging during the follow-up period is to be repeated every 9 weeks or 12 weeks or at the discretion of the attending physician for subjects who discontinue trial treatment for reasons other than disease progression documented disease progression, the start of new anti-cancer treatment, withdrawal of consent, death, or the end of the study, whichever occurs first.

### 7.1.2.6 Tumor Tissue Collection and Correlative Studies Blood Sampling

### 7.1.2.6.1 Tumor Tissue Collection

Mandatory tumor tissue (archival or newly obtained lesion) is required at screening. If archival tissue is not available, a newly obtained core or excisional biopsy of a tumor lesion will be obtained. The screening biopsy must be newly-obtained, which is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Tumor lesions not previously irradiated must be provided (tumors progressing in a prior site of radiation are allowed for PD-L1 characterization). PD-L1 characterization is not required prior to Cycle 1 Day 1. The PD-L1 characterization will be performed retrospectively.

Tumor tissue will be obtained pre- treatment (baseline), between C1D15 and C1D21, and at progression (if patient had complete response (CR), partial response (PR) or stable disease

Product: MK-3475

55 27Jan2022 Protocol/Amendment No.: Version 17/ MDACC#2015-0948

(SD) > 27 weeks) provided there is technically biopsiable tumor, and it is safe for patient to undergo biopsy.

Core needle biopsies should be performed utilizing an 18 gauge needle or thicker whenever feasible or as directed by institutional standards. It is recommended that a minimum of 3 and up to 5 passes are required to ensure adequate tissue is obtained. Alternative biopsy procedures (e.g. cup, punch, excisional, incisional) that are expected to produce a tissue sample greater to or equal than a core biopsy with an 18 gauge core biopsies will also be acceptable. Four fine needle aspirates (FNAs) will also be obtained when feasible for additional exploratory molecular analysis (DNA, RNA, protein). The biopsy approach, number and size may be modified as needed based on tumor size and accessibility.

At screening, archived or newly obtained FFPE (formalin-fixed paraffin embedded) for 5 unstained (4 or 5 micron, 4 micron preferred) slides must be submitted for characterization at a central lab for PD-L1 characterization.

A fine needle aspirate, frozen sample, plastic embedded sample, cell block, clot, bone, bone marrow, cytologic specimen or formalin fixed samples frozen at any point will not be acceptable for IHC analysis. These samples will be sent to a central laboratory at Merck.

### 7.1.2.6.2 Correlative Studies Blood Sampling

Peripheral blood mononuclear cell (PBMC) will be collected at baseline, tumor restaging, in conjunction with biopsies, and time of progression (if patients have had CR/PR/or SD for > 27 weeks). PBMC collections at tumor restaging and in conjunction with biopsies will have a +/-1 day window. Up to six (6) Cell Preparation Tubes (CPT) will be collected at each time point. These samples will be analyzed for the NanoString assay that will evaluate immune-related gene expression signatures and using RNA sequencing, HD peptide analyses, autoantibody profiling analyses and other correlative studies to characterize the molecular phenotype of the tumor and the tumor microenvironment, which have the potential to predict benefit from pembrolizumab.

If subjects are retreated per Section 7.1.5.5, then the PBMC schedule in Section 6.1 will be followed.

Blood samples obtained at baseline or any time point will be used for germline DNA analysis. The analysis of next generation sequencing data for DNA somatic mutations is optimal when germline data is available to ensure that mutation calling is for somatic alterations.

### 7.1.2.7 Tumor Imaging for Correlative Studies

The correlative study imaging will incorporate the standard CT scan parameters or, in the case of MRI, the conventional MRI (T1 pre and post-contrast images, T2-weighted images (T2WI), Fluid attenuating inversion recovery (FLAIR) images) and other standard sequences routinely used. In the case of GBM tumors, additional advanced MRI (MR perfusion [dynamic susceptibility contrast (DSC), dynamic contrast enhancement (DCE) and arterial spin labeling

Product: MK-3475


56

(ASL)], MR- diffusion, and MR spectroscopy) sequences will be obtained. The CT or MRI tumor scans from tumor assessments at baseline, every 9 or 12 weeks (restaging), and at the end-of-treatment will be utilized for these correlative studies. Additional scans or time points will not be required. Imaging post-processing will include but not be limited to RECIST v1.1, irRECIST, advanced quantitative imaging and volume tumor metrics, and voxel-by-voxel radiome sequencing (texture, heterogeneity, energy, etc) imaging analysis. Image analyses will include non-invasive assessments of cell death (apoptosis), active tumor proliferation, tumor invasion, tumor density, vascularity, vascular permeability, microvascular density and metabolite profiles. Exploratory analyses will utilize quantitative imaging tumor metrics and radiome sequencing for texture maps to assess gene signatures of tumor cell apoptosis, invasion and immune cell infiltration. Exploratory analysis using quantitative imaging tumor metrics and texture maps will also be used to assess pseudoprogression, progression and response. These analyses will be compared to a retrospective cohort of patients that have been dichotomously analyzed for lack of inflammatory response versus robust intratumoral inflammatory responses to prospectively validate the sensitivity and specificity of this approach.

### 7.1.2.8 Serial Mutation Assessment

Patients enrolled on this study will be approached for co-enrollment on PA11-0852 Clearinghouse protocol for germline testing for the MD Anderson Cancer Center Personalized Cancer Therapy Program. We expect most patients enrolled will have had hot spot mutation testing or targeted exome profiling performed through the Clearinghouse protocol. If evidence of clinical activity is seen, targeted exome sequencing on a 200-400 gene platform or larger will be performed in patients with objective responses and prolonged stable disease > 27 weeks as well as any patients with rapid progression (this would be done as part of a Institute of Personalized Cancer Therapy Unusual Responder Program. In addition patients who have a mixed response of response with subsequent progression will be approached for optional biopsies for molecular characterization as well as generation of patient-derived xenografts and conditionally-reprogrammed cells. This evaluation will determine the evolution of the mutation and will facilitate functional characterization. Plasma mutations may be assessed with digital PCR or next generation sequencing.

As per the PA11-0852 Clearinghouse protocol, the optional tumor biopsies from baseline and the time of progression (if progression after response or unexpected rapid progression) will be analyzed. Development of new mutations or reversal of the mutations will be analyzed and correlated with clinical response. This will be our exploratory objective and no formal statistical analysis will be done.

#### 7.1.2.9 Microbiome Assessment

### 7.1.2.9.1 Skin Microbiome

Samples will be obtained for skin microbiome testing. Samples may be collected at baseline, at onset of toxicity, and time of tumor restaging. For dermatologic toxicity, samples will be

Product: MK-3475

57 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

obtained from normal tissue and from area of dermatitis (or inflamed skin condition), samples will be obtained from normal tissue and from area of resolved dermatitis (or inflamed skin condition). Up to 11 samples (for culture and DNA) may be collected at each time point. In cases where dermatitis (or inflamed skin condition) occurs in regions that are not designated for skin sample collection, additional skin swab samples may be collected on a case by case basis. Per the laboratory manual, one sample will be used for environmental control.

Patients will be advised to cleanse with only non-antibacterial cleansers during the 7 days before sample collection. To maximize microbial load, no bathing, shampooing or moisturizing will be advised within 24 hours of sample collection, which previously observed produces no discernible shifts in the overall diversity and structures of skin communities. Collection and shipping procedures will be described in the laboratory manual.

Clinical data regarding personal history of atopic dermatitis, family history of atopic dermatitis, current use of topical or antibiotics and date of initiation, past use (within one month) of oral antibiotics with start and end dates, time of last shower, use of antibacterial soap, history of Accutane usage with start and end dates, and history of topical retinoid usage with start and end dates, will be collected.

De-identified samples and de-identified clinical data will be sent to Jackson Laboratory (Julia Oh, PhD) for analyses. The de-identified clinical data will be coded to the samples. The code will only be available to the PI and MDACC study team. Analyzed patient data will be returned to this trial, 2015-0948.

### 7.1.2.9.2 Gut Microbiome

In order to evaluate the gut microbiome, fecal samples will be collected from patients at baseline, onset of toxicity, time of tumor restaging, and End of Treatment visit per the parent treatment protocol.

Sequencing of the V4 region of the 16S bacterial gene will be performed on fecal samples. Whole genome shotgun sequencing may be done on smaller subset of samples on the extreme (e.g. best and worst responders, most toxic vs least toxic). As an initial assessment of microbiome samples; richness, evenness and  $\alpha$ -diversity will be assessed. Alpha-diversity is measure of intra-sample diversity and will be reported as a continuous variable that is calculated based the number and distribution of operational taxonomic units (OTUs refers to classification of microbes into phylum, genus, species, etc.). Indices such as Chao1, Simpson, and Shannon will be used for the determination of alpha-diversity.

Beta-diversity is a measure of inter-sample diversity and will be assessed by the UniFrac method, which calculates the phylogenetic distance between communities. UniFrac distances will be calculated in a weighted or unweighted fashion based on presence or absence of OTUs. In the weighted strategy, the bacterial taxa that are more abundant will get the higher weight.

Product: MK-3475

58 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

Sequencing reads that result in OTU classification will be normalized across the entire dataset by determining the point at which the variance in observed unique OTUs reaches a constant value independent of the sequencing depth. These OTUs will be used determine the relative abundances of bacterial taxa within a sample.

Only de-identified samples will be sent to Jackson Laboratory (Julia Oh, PhD) for analyses. Analyzed patient data will be returned to this trial, 2015-0948.

#### 7.1.2.9.3 Oral Microbiome

Samples will be obtained for oral microbiome testing. Samples will be collected at baseline, at onset of toxicity, and time of tumor restaging. For oral toxicity, samples will be obtained at onset. Collection and shipping procedures will be described in the laboratory manual.

Only de-identified samples will be sent to Jackson Laboratory (Julia Oh, PhD) for analyses. Analyzed patient data will be returned to this trial, 2015-0948.

### 7.1.2.10 Patient-Reported Outcomes

Patient-reported outcomes (PROs) will be collected using select PRO-CTCAE items. Patients will have the baseline PRO-CTCAE completed in clinic on paper. At baseline, patients will specify the preference of delivery of subsequent questionnaires on study- computerized, telephone-based interactive voice response (IVR) system at the patient's preferred time and days of the week or electronically through web-based platforms with RedCap (Research Electronic Data Capture) via an email push.

Subsequent PRO-CTCAE questionnaires will be issued weekly for the first 9 weeks, every 2 weeks until week 54, and every 4 weeks thereafter until End of Treatment or up to Week 81. All questionnaires will have a +/- 2 day window. Questionnaires will be completed at each time point if the patient can be contacted and is willing and able to complete.

### 7.1.2.10.1 PRO Electronic Data Collection and Storage

Symptom data may be collected and managed using REDCap electronic data capture tools hosted at MD Anderson. REDCap (www.project-redcap.org) is a secure, web-based application with controlled access designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless downloads to common statistical packages; and 4) procedures for importing data from external sources.

REDCap (https://redcap.mdanderson.org) is hosted on a secure server by MD Anderson Cancer Center's Department of Research Information Systems & Technology Services. REDCap has undergone a Governance Risk & Compliance Assessment (05/14/14) by MD

Product: MK-3475


59

Anderson's Information Security Office and found to be compliant with HIPAA, Texas Administrative Codes 202-203, University of Texas Policy 165, federal regulations outlined in 21CFR Part 11, and UTMDACC Institutional Policy #ADM0335. Those having access to the data file include the study PI and research team personnel. Users are authenticated against MDACC's Active Directory system. External collaborators are given access to projects once approved by the project sponsor. The application is accessed through Secure Socket Layer (SSL).

All protected health information (PHI) will be removed from the data when it is exported from REDCap for analysis. All dates for a given patient will be shifted by a randomly generated number between 0 and 364, thus preserving the distance between dates. Dates for each patient will be shifted by a different randomly generated number. After publication, study data will be archived in REDCap.

### 7.1.2.10.2 IVR system

We will use paper or a secure electronic method when the patient is in the clinic, and use an interactive voice response (IVR) system, phone calls by field coordinators, secure web access, or regular mail when patients are away from the clinic. The method of collecting the PRO-CTCAE assessments will be based on patient preference and may be varied throughout the study based on patient request. An IVR system can greatly facilitate the longitudinal tracking of symptoms in patients. IVR systems are programmed to call patients at home for symptom assessment. The IVR system asks patients to rate each symptom and interference item on the PRO-CTCAE numeric scales using the keypad of a touchtone telephone.

Participants electing to use the IVR system may be provided with an informational brochure outlining the steps to complete an IVR call. A telephone number will be provided in the event of questions or problems. Patients will also be given a Patient Identification Number (PIN) for access to the system. IVR calls will be scheduled at a time that is convenient for the patient.

Completion or failure of calls will be monitored by the research staff. In the event of missed calls, a notification screen will appear in the IVR system to alert the research staff. The research staff will then contact the patient, check on their status and, if possible, complete the assessment with the patient during the telephone interview. The system will continue calling the patient at the preset schedule.

The IVR symptom and interference data will be available on an MD Anderson intranet site with access limited to authorized project staff only. Patient data will be identified by subject study number.

Product: MK-3475 60 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

# 7.1.3 Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below. Laboratory tests for hematology, chemistry, urinalysis, and others are specified in Table 7.

Product: MK-3475 61 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

**Table 7 Laboratory Tests** 

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hematocrit | Albumin | Blood | Serum β-human chorionic gonadotropin† |
| Hemoglobin | Alkaline phosphatase | Glucose | (β-hCG)† |
| Platelet count | Alanine aminotransferase (ALT) | Protein | PT (INR) |
| WBC (total and differential) | Aspartate aminotransferase (AST) | Specific gravity | aPTT |
| Red Blood Cell Count | Lactate dehydrogenase (LDH) | Microscopic exam (If abnormal) | Total thriiodothyronine (T3) |
| Absolute Neutrophil Count | Carbon Dioxide ‡ | results are noted | Free thyroxine (T4) |
| Absolute Lymphocyte Count | (CO <sub>2</sub> or biocarbonate) | Urine pregnancy test † | Thyroid stimulating hormone (TSH) |
| | Uric Acid | | |
| | Calcium | | |
| | Chloride | | Blood for correlative studies |
| | Glucose | | |
| | Phosphorus | | |
| | Potassium | | |
| | Sodium | | |
| | Magnesium | | |
| | Total Bilirubin | | |
| | Direct Bilirubin (If total bilirubin is elevated above the upper limit of normal) | | |
| | Total protein | | |
| | Blood Urea Nitrogen | | |

<sup>†</sup> Perform on women of childbearing potential only. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test will be required.

<sup>‡</sup> If considered standard of care in your region.

Product: MK-3475

62 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

Laboratory tests for screening or entry into the Second Course Phase should be performed within 28 days prior to the first dose of treatment. After Cycle 1, pre-dose laboratory procedures can be conducted up to 72 hours (3 days) prior to each dosing on Day 1 of each subsequent cycle. Results must be reviewed by the investigator or qualified designee and found to be acceptable prior to each dose of trial treatment.

#### 7.1.4 Other Procedures

#### 7.1.4.1 Withdrawal/Discontinuation

When a subject discontinues/withdraws prior to trial completion, all applicable activities scheduled for the final trial visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 - Assessing and Recording Adverse Events. Subjects who a) attain a CR or b) complete 24 months of treatment with pembrolizumab may discontinue treatment with the option of restarting treatment if they meet the criteria specified in Section 7.1.5.5. After discontinuing treatment following assessment of CR, these subjects should return to the site for a Safety Follow-up Visit (described in Section 7.1.5.3) and then proceed to the Follow-Up Period of the study (described in Section 7.1.5.4).

If a patient withdraws consent for further study treatment, the patient should still be followed for progression and survival. If a patient withdraws consent for further participation in the study, follow-up assessments will be discontinued.

### 7.1.4.2 Blinding/Unblinding

This is an open label trial; there is no blinding for this trial.

### 7.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

### 7.1.5.1 Screening Period

Approximately 28 days prior to enrollment, potential subjects will be evaluated to determine that they fulfill the entry requirements as set forth in Section 5.1. Visit requirements are outlined in Section 6.0 – Trial Flow Chart.

After providing main study consent, subjects will undergo the screening period. Results of a test performed prior to the subject signing consent as part of routine clinical management are acceptable in lieu of a screening test if performed within the specified time frame. Screening procedures are to be completed within 28 days prior to the first dose of trial treatment except for the following:

Product: MK-3475 63 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

• Laboratory tests are to be performed within 28 days prior to the first dose of trial treatment

- For women of reproductive potential, a urine pregnancy test will be performed within 72 hours (3 days) prior to the first dose of trial treatment. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy test will be required (performed by the local study site laboratory)
- Archival tissue collection for PD-L1 characterization are not required to be completed within 28 days prior to the first dose of trial treatment

Subjects may be rescreened after initially failing to meet the inclusion/exclusion criteria. Results from assessments performed during the initial screening period are acceptable in lieu of a repeat screening test if performed within the specified time frame and the inclusion/exclusion criteria is met.

#### 7.1.5.2 Treatment Period

Visit requirements are outlined in <u>Section 6.0</u> – Trial Flow Chart.

#### 7.1.5.3 Post-Treatment Visits

# 7.1.5.3.1 Safety Follow-Up Visit

The mandatory Safety Follow-Up Visit should be conducted approximately 30 days ( $\pm$  7 days) after the last dose of trial treatment or before the initiation of a new anti-cancer treatment, whichever comes first. All AEs that occur prior to the Safety Follow-Up Visit should be recorded. Subjects with an AE of Grade > 1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anti-neoplastic therapy, whichever occurs first. SAEs that occur within 90 days of the end of treatment or before initiation of a new anti-cancer treatment should also be followed and recorded. Subjects who are eligible for retreatment with pembrolizumab (as described in Section 7.1.5.5) may have up to two safety follow-up visits, one after the Treatment Period and one after the Second Course Phase.

### 7.1.5.4 Follow-up Visits

Subjects who discontinue trial treatment for a reason other than disease progression will move into the Follow-Up Phase. Post discontinuation, subjects will be assessed every 9 weeks, 12 weeks, or at the discretion of the treating physician ( $\pm$  7 days) by radiologic imaging to monitor disease status. Every effort should be made to collect information regarding disease status until the start of new anti-neoplastic therapy, disease progression, death, end of the study or if the subject begins retreatment with pembrolizumab as detailed in Section 7.1.5.5. Information regarding post-study anti-neoplastic treatment will be collected if new treatment is initiated.

Product: MK-3475


Subjects who are eligible to receive retreatment with pembrolizumab according to the criteria in <u>Section 7.1.5.5</u> will move from the follow-up phase to the Second Course Phase when they experience disease progression. Details are provided in <u>Section 6.1</u> – Trial Flow Chart for Retreatment.

### 7.1.5.4.1 Survival Follow-up

Once a subject experiences confirmed disease progression or starts a new anti-cancer therapy, the subject moves into the survival follow-up phase, and survival data will be collected from a chart review, patient visit, or by telephone every 12 weeks ( $\pm$  4 weeks) to assess for survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.

### 7.1.5.5 Second Course Phase (Retreatment Period)

Subjects who stop pembrolizumab with SD or better may be eligible for up to one year of additional pembrolizumab therapy if they progress after stopping study treatment. This retreatment is termed the Second Course Phase of this study and is only available if the study remains open and the subject meets the following conditions:

#### • Either

- Stopped initial treatment with pembrolizumab after attaining an investigatordetermined confirmed CR according to RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated, and
  - Was treated for at least 27 weeks (9 cycles) with pembrolizumab before discontinuing therapy
  - Received at least two treatments with pembrolizumab beyond the date when the initial CR was declared

#### OR

o Had SD, PR or CR and stopped pembrolizumab treatment after 24 months of study therapy for reasons other than disease progression or intolerability

### AND

- Experienced an investigator-determined confirmed radiographic disease progression after stopping their initial treatment with pembrolizumab
- Did not receive any anti-cancer treatment since the last dose of pembrolizumab
- Has a performance status of 0 or 1 on the ECOG Performance Scale

Product: MK-3475 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

65

Demonstrates adequate organ function as detailed in Section 5.1.2

- Female subject of childbearing potential should have a negative serum or urine pregnancy test within 72 hours prior to receiving retreatment with study medication.
- Female subject of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of child bearing potential are those who have not been surgically sterilized or have been free from menses for > 1 year.
- Male subject should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
- Does not have a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the trial or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Subjects who restart treatment will be retreated at the same dose and dose interval as when they last received pembrolizumab. Treatment will be administered for up to one additional year.

Visit requirements are outlined in Section 6.1 – Trial Flow Chart.

#### 7.2 **Assessing and Recording Adverse Events**

An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocolspecified procedure, whether or not considered related to the medicinal product or protocolspecified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Merck's product, is also an adverse event.

Changes resulting from normal growth and development that do not vary significantly in frequency or severity from expected levels are not to be considered adverse events. Examples of this may include, but are not limited to, teething, typical crying in infants and children and onset of menses or menopause occurring at a physiologically appropriate time.

Merck product includes any pharmaceutical product, biological product, device, diagnostic agent or protocol-specified procedure, whether investigational (including placebo or active

Product: MK-3475

66 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

comparator medication) or marketed, manufactured by, licensed by, provided by or distributed by Merck for human use.

Adverse events may occur during the course of the use of Merck product in clinical trials or within the follow-up period specified by the protocol, or prescribed in clinical practice, from overdose (whether accidental or intentional), from abuse and from withdrawal.

Adverse events may also occur in screened subjects during any pre-allocation baseline period as a result of a protocol-specified intervention, including washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

Progression of the cancer under study is not considered an adverse event unless it is considered to be drug related by the investigator.

All adverse events will be recorded from the time the consent form is signed through 30 days following cessation of treatment and at each examination on the Adverse Event case report forms/worksheets. The reporting timeframe for adverse events meeting any serious criteria is described in section 7.2.3.1.

The study drug-related adverse event data will be collected and stored in the Investigational Cancer Therapeutics database, Molecular and Clinical Data Integrated Platform (MOCLIP). The PI or designee will be responsible for determining attribution for all events, and this will be documented in the electronic medical record.

# 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the **IND Sponsor and to Merck**

For purposes of this trial, an overdose of pembrolizumab will be defined as any dose of 1,000 mg or greater (≥5 times the indicated dose). No specific information is available on the treatment of overdose of pembrolizumab. Appropriate supportive treatment should be provided if clinically indicated. In the event of overdose, the subject should be observed closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated.

If an adverse event(s) is associated with ("results from") the overdose of a Merck product, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.

If a dose of Merck's product meeting the protocol definition of overdose is taken without any associated clinical symptoms or abnormal laboratory results, the overdose is reported as a nonserious Event of Clinical Interest (ECI), using the terminology "accidental or intentional overdose without adverse effect."

Product: MK-3475


67

All reports of overdose with and without an adverse event must be reported within 24 hours to the IND Sponsor and within 2 working days hours to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

### 7.2.2 Reporting of Pregnancy and Lactation to the IND Sponsor and to Merck

Although pregnancy and lactation are not considered adverse events, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject (spontaneously reported to them), including the pregnancy of a male subject's female partner that occurs during the trial or within 120 days of completing the trial completing the trial, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier. All subjects and female partners of male subjects who become pregnant must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

Such events must be reported within 24 hours to the IND Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

### 7.2.3 Immediate Reporting of Adverse Events to the IND Sponsor and to Merck

#### 7.2.3.1 Serious Adverse Events

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or the sponsor, it results in any of the following outcomes:

- Death
- A life-threatening adverse drug experience any adverse experience that places the patient, in the view of the initial reporter, at immediate risk of death from the adverse experience as it occurred. It does not include an adverse experience that, had it occurred in a more severe form, might have caused death.
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- A congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse (21 CFR 312.32).

Product: MK-3475 68 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

• Important medical events as defined above, may also be considered serious adverse events. Any important medical event can and should be reported as an SAE if deemed appropriate by the Principal Investigator or the IND Sponsor, IND Office.

- All events occurring during the conduct of a protocol and meeting the definition of a
  SAE must be reported to the IRB in accordance with the timeframes and procedures
  outlined in "The University of Texas M. D. Anderson Cancer Center Institutional
  Review Board Policy for Investigators on Reporting Unanticipated Adverse Events for
  Drugs and Devices". Unless stated otherwise in the protocol, all SAEs, expected or
  unexpected, must be reported to the IND Office, regardless of attribution (within 5
  working days of knowledge of the event).
- All life-threatening or fatal events, that are unexpected, and related to the study drug, must have a written report submitted within 24 hours (next working day) of knowledge of the event to the Safety Project Manager in the IND Office.
- Unless otherwise noted, the electronic SAE application (eSAE) will be utilized for safety reporting to the IND Office and MDACC IRB.
- Serious adverse events will be captured from the time of the first protocol-specific intervention, until 90 days after the last dose of drug, unless the participant withdraws consent. Serious adverse events must be followed until clinical recovery is complete and laboratory tests have returned to baseline, progression of the event has stabilized, or there has been acceptable resolution of the event.
- Additionally, any serious adverse events that occur after the 90 day time period that are related to the study treatment must be reported to the IND Office. This may include the development of a secondary malignancy.

### **Reporting to FDA:**

• Serious adverse events will be forwarded to FDA by the IND Sponsor (Safety Project Manager IND Office) according to 21 CFR 312.32.

It is the responsibility of the PI and the research team to ensure serious adverse events are reported according to the Code of Federal Regulations, Good Clinical Practices, the protocol guidelines, the sponsor's guidelines, and Institutional Review Board policy.

Any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study that occurs to any subject from the time the consent is signed through 90 days following cessation of treatment, or the initiation of new anti-cancer therapy, whichever is earlier, whether or not related to Merck product, must be reported within 2 working days to Merck Global Safety.

Additionally, any serious adverse event, considered by an investigator who is a qualified physician to be related to Merck product that is brought to the attention of the investigator at any time following consent through the end of the specified safety follow-up period specified

Product: MK-3475


69

in the paragraph above, or at any time outside of the time period specified in the previous paragraph also must be reported immediately to the IND Sponsor and to Merck.

# SAE reports and any other relevant safety information are to be forwarded to the Merck Global Safety facsimile number: +1-215-993-1220

A copy of all 15 Day Reports and Annual Progress Reports is submitted as required by FDA, European Union (EU), Pharmaceutical and Medical Devices agency (PMDA) or other local regulators. Investigators will cross reference this submission according to local regulations to the Merck Investigational Compound Number (IND, CSA, etc.) at the time of submission. Additionally investigators will submit a copy of these reports to Merck & Co., Inc. (Attn: Worldwide Product Safety; FAX 215 993-1220) at the time of submission to FDA.

All subjects with serious adverse events must be followed up for outcome.

#### 7.2.3.2 Events of Clinical Interest

Selected non-serious and serious adverse events are also known as Events of Clinical Interest (ECI) and must be recorded as such on the Adverse Event case report forms/worksheets and reported within 24 hours to the IND Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220).

For the time period beginning when the consent form is signed until treatment, any ECI, or follow up to an ECI, that occurs to any subject must be reported within 24 hours to the IND Sponsor and within 2 working days to Merck Global Safety if it causes the subject to be excluded from the trial, or is the result of a protocol-specified intervention, including but not limited to washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

For the time period beginning at treatment through 90 days following cessation of treatment, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier, any ECI, or follow up to an ECI, whether or not related to Merck product, must be reported within 24 hours to the IND Sponsor and within 24 hours to Merck Global Safety.

Events of clinical interest for this trial include:

- 1. An overdose of Merck product, as defined in <u>Section 7.2.1</u> Definition of an Overdose for This Protocol and Reporting of Overdose to the IND Sponsor, that is not associated with clinical symptoms or abnormal laboratory results.
- 2. An elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing.\*

Product: MK-3475

70 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

\*Note: These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology. This is a recommendation; however, the clinical decision will be made by the PI and consulting/treating physician.

### 7.2.3.3 Protocol-Specific Exceptions to Serious Adverse Event Reporting

Efficacy endpoints as outlined in this section will not be reported to Merck as described in Section 7.2.3- Immediate Reporting of Adverse Events to the IND Sponsor and to Merck, unless there is evidence suggesting a causal relationship between the drug and the event. Any such event will be submitted to the IND Sponsor within 24 hours and to Merck Global Safety within 2 working days either by electronic or paper media.

Specifically, the suspected/actual events covered in this exception include any event that is disease progression of the cancer under study.

The IND Sponsor will monitor unblinded aggregated efficacy endpoint events and safety data to ensure the safety of the subjects in the trial. Any suspected endpoint which upon review is not progression of the cancer under study will be forwarded to Merck Global Safety as a SAE within 2 working days of determination that the event is not progression of the cancer under study

Hospitalization related to convenience (e.g. transportation issues etc.) will not be considered a SAE.

### 7.2.4 Evaluating Adverse Events

An investigator who is a qualified physician will evaluate all adverse events according to the NCI Common Terminology for Adverse Events (CTCAE), version 4.03. Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded on the adverse event case report forms/worksheets.

All adverse events regardless of CTCAE grade must also be evaluated for seriousness.

Product: MK-3475 71 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

# **Table 8 Evaluating Adverse Events**

An investigator who is a qualified physician, will evaluate all adverse events as to:

| V4.03 CTCAE<br>Grading | Grade 1 | Mild; asymptomatic or mid symptoms; clinical or diagnostic observations only; intervention not indicated. |
|---|---|---|
| | Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. |
| | Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation or hospitalization indicated; |
| | | disabling; limiting self-care ADL. |
| | Grade 4 | Life threatening consequences; urgent intervention indicated. |
| | Grade 5 | Death related to AE |
| Seriousness | A serious adverse e | event is any adverse event occurring at any dose or during any use of Merck product that: |
| | †Results in death; | |
| | | g; or places the subject, in the view of the investigator, at immediate risk of death from the event as it occurred (Note: This does not include an |
| | | had it occurred in a more severe form, might have caused death.); or |
| | | istent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions); or |
| | | longs an existing inpatient hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay, even if the |
| | | precautionary measure for continued observation. (Note: Hospitalization [including hospitalization for an elective procedure] for a preexisting |
| | | s not worsened does not constitute a serious adverse event.); or |
| | | nomaly/birth defect (in offspring of subject taking the product regardless of time to diagnosis);or |
| | | that is not a condition of the study) or |
| | | nether accidental or intentional). Any adverse event associated with an overdose is considered a serious adverse event. An overdose that is not |
| | | adverse event is considered a non-serious event of clinical interest and must be reported within 24 hours. |
| | | medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, |
| | | riate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes |
| | | lesignated above by a †). |
| Duration | | d stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units |
| Action taken | | ent cause the Merck product to be discontinued? |
| Relationship to | | duct cause the adverse event? The determination of the likelihood that the Merck product caused the adverse event will be provided by an |
| test drug | | a qualified physician. The investigator's signed/dated initials on the source document or worksheet that supports the causality noted on the AE |
| | | a medically qualified assessment of causality was done. This initialed document must be retained for the required regulatory time frame. The |
| | | ntended as reference guidelines to assist the investigator in assessing the likelihood of a relationship between the test drug and the adverse event |
| | based upon the ava | |
| | | nponents are to be used to assess the relationship between the Merck product and the AE; the greater the correlation with the components and |
| | | ments (in number and/or intensity), the more likely the Merck product caused the adverse event (AE): |
| | Exposure | Is there evidence that the subject was actually exposed to the Merck product such as: reliable history, acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or measurement of drug/metabolite in bodily specimen? |
| | Time Course | Did the AE follow in a reasonable temporal sequence from administration of the Merck product? |
| | | Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with investigational medicinal product)? |
| | Likely Cause | Is the AE not reasonably explained by another etiology such as underlying disease, other drug(s) vaccine(s), or other host or environmental factors |

Product: MK-3475 72 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

| Was the Merck product (continued) Rechallenge Rechallenge Rechallenge Rechallenge Rechallenge Rechallenge Rechallenge Re | |
|---|---|
| Continued If yes, this is a positive dechallenge. If no, this is a negative dechallenge. (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE of the Merck product; or (3) the trial is a single-dose drug trial); or (4) Merck product(s) is/are only used to the Merck product in this study? Rechallenge | |
| (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the AE rof the Merck product; or (3) the trial is a single-dose drug trial); or (4) Merck product(s) is/are only used to the Merck product in this study? If yes, did the AE recur or worsen? If yes, this is a positive rechallenge. If no, this is a negative rechallenge. (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) (3) Merck product(s) is/are used only one time). NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. State clinical/pathological presentation of the AE consistent with previous knowledge regarding the Mer or toxicology? The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Ves, there is a reasonable possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the is reasonable. The AE is more likely explained by the Merck product than by another cause. | |
| Rechallenge Rechallenge Was the subject re-exposed to the Merck product in this study? If yes, did the AE recur or worsen? If yes, this is a positive rechallenge. If no, this is a negative rechallenge. (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) (3) Merck product(s) is/are used only one time). NOTE: If A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the is reasonable. The AE is more likely explained by the Merck product than by another cause. | |
| Was the subject re-exposed to the Merck product in this study? If yes, did the AE recur or worsen? If yes, did the AE recur or worsen? If yes, this is a positive rechallenge. If no, this is a negative rechallenge. (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) (3) Merck product(s) is/are used only one time). NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Mer or toxicology? Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Mer or toxicology? Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a stream of the following scale of criteria as guidance (not all criteria must be present to be indicative of a stream of the possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the relationship. The AE is more likely explained by the Merck product than by another cause. | |
| If yes, did the AE recur or worsen? If yes, this is a positive rechallenge. If no, this is a negative rechallenge. (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) (3) Merck product(s) is/are used only one time). NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Mer or toxicology? The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the relationship. | one time.) |
| If yes, this is a positive rechallenge. If no, this is a negative rechallenge. (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) (3) Merck product(s) is/are used only one time). NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Monitory of the AE is more likely explained by the Merck product than by another cause. | |
| (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, or (2) (3) Merck product(s) is/are used only one time). NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to Profile to the showe elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the seasonable is reasonable. The AE is more likely explained by the Merck product than by another cause. | |
| (3) Merck product(s) is/are used only one time). NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Meror toxicology? The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Merck product to the Merck product. The temporal sequence of the AE onset relative to the possibility of Merck product There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the possibility of Merck product There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the possibility of Merck product. The temporal sequence of the AE onset relative to the Merck product than by another cause. | |
| NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS SERIOUS A CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Mer or toxicology? The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the sequence of the AE onset relative to | the trial is a single-dose drug trial); or |
| CAUSED BY THE MERCK PRODUCT, OR IF REEXPOSURE TO THE MERCK PRODUCT POSES SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a March Product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the is reasonable. The AE is more likely explained by the Merck product than by another cause. | ND WHICH MAN HAVE DEEN |
| SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED IN A MONITOR AS PER DOSE MODIFICATION GUIDELINES IN THE PROTOCOL. Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to a consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a fine possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the is reasonable. The AE is more likely explained by the Merck product than by another cause. | |
| Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Yes, there is a reasonable possibility of Merck product relationship. The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. There is evidence of criteria as guidance (not all criteria must be present to be indicative of a finite possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the possibility of Merck product relationship. | |
| Consistency with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to a consideration of the above elements. Record one of the following Ves, there is a reasonable possibility of Merck product relationship. Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Merck product with previous knowledge regarding the Merck profile. Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Merck profile. In the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Merck profile. In the clinical/pathological presentation of the AE consistent with previous knowledge regarding the Merck profile. | DVANCE BY THE U.S. CLINICAL |
| with Trial Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Ves, there is a reasonable possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the is reasonable. The AE is more likely explained by the Merck product than by another cause. | . 1 1 1 1 |
| Treatment Profile The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to a consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a March product is reasonable in relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the more likely explained by the Merck product than by another cause. | ck product of drug crass pharmacology |
| The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Market product of the AE onset relative to the Merck product. The temporal sequence of the AE onset relative to the Merck product than by another cause. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the Merck product than by another cause. | |
| The assessment of relationship will be reported on the case report forms /worksheets by an investigator who is a qualified physician according to be consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a Market product. The temporal sequence of the AE onset relative to the possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the merck product than by another cause. | |
| Consideration of the above elements. Record one of the following Use the following scale of criteria as guidance (not all criteria must be present to be indicative of a March possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the Merck product than by another cause. | nis/her best clinical judgment, including |
| Yes, there is a reasonable possibility of Merck product relationship. There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative to the Merck product than by another cause. | |
| possibility of Merck product is reasonable. The AE is more likely explained by the Merck product than by another cause. | Merck product relationship). |
| No, there is not a reasonable Subject did not receive the Merck product OR temporal sequence of the AE onset relative to administration | he administration of the Merck product |
| No, there is not a reasonable Subject did not receive the Merck product OR temporal sequence of the AE onset relative to administration | |
| possibility Merck product relationship OR there is another obvious cause of the AE. (Also entered for a subject with overdose without an associated and the control of the AE.) | |

73

### 7.2.5 Sponsor Responsibility for Reporting Adverse Events

All Adverse Events will be reported to regulatory authorities, IRB/IECs and investigators in accordance with all applicable global laws and regulations.

#### 8.0 STATISTICAL ANALYSIS PLAN

This section outlines the statistical analysis strategy and procedures for the study. If, after the study has begun, changes are made to primary and/or key secondary hypotheses, or the statistical methods related to those hypotheses, then the protocol will be amended (consistent with ICH Guideline E-9).

#### **Statistical Analysis Plan Summary** 8.1

This section contains a brief summary of the statistical analyses for this trial. There will be 10 cohorts included in the overall population of different cancer types. All patients who have received at least 1 dose of study medication with at least one adequate on-study tumor assessment will be included in the efficacy analysis. If a patient discontinued the study before the first radiological assessment due to progression of disease, either radiological or clinical, they will be considered evaluable and will be included in the efficacy analysis. However, if the patient discontinued the study before 27 weeks due to reasons other than progression of disease or death, they will be considered non evaluable for assessment of primary efficacy endpoint (alive and progression-free at 27 weeks). All patients who received at least 1 dose of study medication will be considered for the toxicity analysis.

### 8.1.1 General Analyses

Tabulations will be produced for appropriate demographic, baseline, efficacy and safety parameters. For categorical variables, summary tabulations of the number and percentage of subjects within each category (with a category for missing data) of the parameter will be presented, as well as two-sided 95% confidence intervals, unless otherwise stated. For continuous variables, the number of subjects, mean, median, standard deviation (SD), minimum, and maximum values will be presented. Time-to-event data will be summarized using Kaplan-Meier methodology using 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals, as well as percentage of censored observations.

### 8.1.2 Efficacy Analyses

Clinical efficacy will be measured by non-progression rate (NPR) at 27 weeks as defined as the percentage of patients who are alive and progression-free at 27 weeks as assessed by RECIST v1.1 criteria or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated. A 95% confidence interval of response rate will be estimated based on a binomial distribution. Other efficacy parameters such as percentage of

Product: MK-3475


74

patients with objective response, clinical benefit (CR, PR, SD >/=4 months), PFS, OS and DOR and their correlation to PD-L1 status will also be analyzed.

### 8.1.3 Safety Analysis

For the objective of describing the toxicity profile, descriptive statistics will be provided on the grade and type of toxicity by dose level.

#### 8.1.3.1 Adverse Events

Adverse Events (AEs) will be coded using the NCI-CTCAE (4.03) dictionary and displayed for all study patients combined. Analyses of AEs will be performed for those events that are considered treatment emergent, where treatment-emergent is defined as any AE with onset or worsening of a pre-existing condition on or after the first administration of study medication through 30 days following last dose or any event considered drug-related by the investigator through the end of the study. AEs with partial dates will be assessed using the available date information to determine if treatment-emergent; AEs with completely missing dates will be assumed to be treatment-emergent.

AEs will be summarized by patient incidence rates, therefore, in any tabulation, a patient contributes only once to the count for a given AE preferred term. The number and percentage of patients with any treatment-emergent AE will be summarized for all study patients combined. The number and percentage of patients with treatment-emergent AEs assessed by the Investigator as at least possibly related to treatment will also be tabulated. The number and percentage of patients with any grade  $\geq 3$  treatment-emergent AE will be tabulated in the same manner. In the event a patient experiences repeated episodes of the same AE, then the event with the highest severity and/or strongest causal relationship to study treatment will be used for purposes of tabulations. Serious AEs will also be tabulated.

No formal hypothesis-testing analysis of AE incidence rates will be performed. All AEs (treatment emergent and post-treatment) will be listed in patient data listings. By-patient listings will be provided for the following: patient deaths; serious AEs; and AEs leading to withdrawal.

#### 8.1.3.2 Laboratory Data

The actual value and change from baseline to each on study evaluation will be summarized for each clinical laboratory parameter, including hematology and clinical chemistry, for all study patients combined. In the event of repeat values, the last non-missing value per study day/time will be used. Severity of select clinical lab measures will be determined using CTCAE criteria (e.g. those measures that have a corresponding CTCAE grade classification). Labs with CTCAE grades greater than or equal to 3 will be presented in a data listing. Shift tables that present changes from baseline to worst on-study values relative to CTCAE classification ranges will be produced.

Product: MK-3475

Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

75

### 8.1.4 Power and Sample Size

The sample size for this study is based on the Simon's optimal two-stage design.<sup>17</sup>

This trial has futility interim analyses for the well-defined expansion cohorts of Cohorts 1-9, and the endpoint is 27-week PFS (referred to as non-progression rate, NPR). Cohorts 1-9 will follow a two-stage design with 12 patients in the first stage and 13 in the second stage. If among the 12 evaluable patients enrolled in the first stage, 3 or more patients are alive and progressionfree at 27 weeks, enrollment into the second stage will begin. If more than 7 of the 25 total evaluable patients in a cohort are alive and progression-free at 27 weeks, the drug will be considered worthy of further study in that cohort. The null success rate is set at 20% and the alternative at 40% for each cohort. This design has a 10% Type I error rate, 82% power and 56% probability of stopping after the first stage if the true 27-week PFS rate is 20%.

The maximum accrual will be 250 patients (25 patients x 10 cohorts). In order to get 250 evaluable patients, up to 275 patients may need to be enrolled.

In Cohort 10, there will not be a two-step design since the cohort will be composed of a heterogeneous tumor population. If one patient of a tumor type experiences success defined as subjects being alive and progression-free at 27 weeks, then that tumor type may be expand to an additional 14 patients.

### 8.1.5 Interim Analyses

For Cohorts 1-9, in accordance with the Simon two-stage study design described in Section 8.1.4, there will be a preliminary assessment of efficacy for each cohort after the first 12 evaluable patients enrolled in that cohort have 27-week data available to assess efficacy. Note that this initial analysis for a cohort may take place sooner than when the 12th patient has available data, should there be 3 or more responders after fewer than 12 patients are enrolled. Should the trial be terminated at the first stage, all efficacy and safety analyses as noted above will be performed. Patient enrollment will be suspended pending observation of the needed numbers of responses.

### **Response Monitoring:**

### STAGE 1:

A Futility Summary will be submitted to the IND Medical Monitor after 12 subjects are evaluable for response (at 27 weeks) per cohort.

#### STAGE 2:

A final Response Summary will be submitted to the IND Medical Monitor after there are 25 evaluable patients for response per cohort.

The final analysis for each cohort will take place after there are 25 patients evaluable for analysis of efficacy. Additional data summarization may take place after all available survival data are collected, or after investigator decision, as appropriate.

76 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

#### 8.2 **Statistical Analysis Plan**

### 8.2.1 Responsibility for Analyses

The statistical analysis of the data obtained from this study will be the responsibility of the University of Texas MD Anderson Cancer Center, Biostatistics department. A detailed analysis plan has been developed and will be implemented.

#### 8.3 **Study Objectives**

### 8.3.1 Primary Objective

**Objective:** To obtain early indication of efficacy by evaluation of non-progression rate (NPR) at 27 weeks as defined as the percentage of patients who are alive and progression-free at 27 weeks, as assessed by RECIST v1.1 or irRECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated in patients with advanced tumor types receiving pembrolizumab.

### 8.3.2 Secondary Objectives

- (1) **Objective**: To correlate efficacy by evaluation of tumor size to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.
- (2) **Objective:** To evaluate safety and tolerability of pembrolizumab in patients with advanced tumors.
- (3) **Objective:** To evaluate the percentage of patients with objective response (CR or PR), clinical benefit (CR, PR, stable disease [SD] >/=4 months), progression free survival (PFS), overall survival (OS), and duration of response (DOR) as assessed by RECIST v1.1 in patients with advanced tumor types receiving pembrolizumab.
- (4) **Objective:** To evaluate the percentage of patients with objective response (CR or PR), clinical benefit (CR, PR, or SD >/=4 months), PFS, and DOR as assessed by irRECIST in patients with advanced tumor types receiving pembrolizumab.
- (5) **Objective:** To correlate the NPR at 27 weeks (9 cycles), objective response (CR or PR), clinical benefit (CR, PR, or SD >/=4 months), PFS, OS, and DOR to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.

### **8.3.3** Exploratory Objectives:

(1) **Objective:** To evaluate the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness in patients with advanced tumor types receiving pembrolizumab.

Product: MK-3475

77 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

(2) **Objective:** To correlate the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.

- (3) **Objective:** To identify imaging characteristics associated with immunological changes in tumor following treatment with pembrolizumab.
- (4) **Objective:** To compare tumor mutation burden and serial assessment of mutation status in biopsies obtained at baseline and progression in patients with advanced tumor types receiving pembrolizumab.
- (5) **Objective:** To evaluate PRO utilizing the NCI PRO-CTCAE items.
- (6) Objective: For patients that experience dermatologic irAEs, to compare the skin microbiome of normal (non-rash) skin to skin microbiome of area with rash.
- (7) **Objective:** For patients that experience oral irAEs, to assess the oral microbiome at baseline, at onset of toxicity, and time of tumor restaging
- (8) **Objective:** For patients that experience gut irAEs, to assess the gut microbiome at baseline, onset of toxicity, time of tumor restaging, and End of Treatment visit per the parent treatment protocol.
- (9) **Objective:** To analyze tumor-infiltrating lymphocytes using H&E stained whole slide images.

#### 8.4 **Hypotheses:**

Intravenous administration of single agent pembrolizumab (MK-3475) to subjects with a given PD-L1 positive advanced tumor type will result in an NPR at 27 weeks greater than 20% based on RECIST v1.1 criteria or irRECIST or according to tumor evaluation criteria best suitable and accepted for the tumor type evaluated.

#### 8.5 **Analysis Endpoints**

Efficacy endpoints will be evaluated as aggregate and between PD-L1 and non-PD-L1 expressing tumor types within and across tumor types.

### 8.5.1.1 Efficacy Endpoints

The primary efficacy endpoint is NPR at 27 weeks, defined as the proportion of subjects in the analysis population who have has no progression of disease by 27 weeks. Response for the primary analysis will be determined by the investigator assessment, and a confirmation assessment is required per RECIST v1.1 or irRECIST or according to tumor evaluation criteria best suitable and accepted for the tumor type evaluated.

Product: MK-3475

78 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

Secondary efficacy endpoints include: objective response (CR, PR); clinical benefit (CR, PR or SD >/=4 months) according to RECIST, v1.1 or irRECIST;; progression-free survival (PFS), defined as the time from allocation to the first documented disease progression according to RECIST v1.1 or irRECIST or death due to any cause, whichever occurs first; and overall survival (OS). The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that progressive disease is objectively documented. The duration of overall complete response is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented. Stable disease is measured from the start of the treatment until the criteria for progression are met.

Per RECIST 1.1 or irRECIST, response should be confirmed by a repeat radiographic assessment not less than 4 weeks from the date the response was first documented. The scan for confirmation of response may be performed at the earliest 4 weeks after the first indication of response, or at the next scheduled scan, whichever is clinically indicated.

Disease progression should be confirmed at least 4 weeks after the first scan indicating progressive disease in clinically stable subjects. Subjects who have unconfirmed disease progression may continue on treatment until progression is confirmed provided they have met the conditions detailed in Section 7.1.2.5. Symptomatic deterioration may indicate progressive disease (PD). However, radiological confirmation of PD is strongly recommended.

#### 8.5.1.2 Safety Endpoints

The primary safety endpoints are AEs graded using CTCAE (Version 4.03) criteria. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received pembrolizumab (MK-3475), including serious adverse events (SAEs), events of clinical interest (ECIs), and immune-related adverse experiences (irAEs). Other safety endpoints include laboratory safety assessments, ECOG performance status, vital signs and physical examinations.

#### **8.5.1.3** Exploratory Endpoints

Image analyses will include non-invasive assessments of cell death (apoptosis), active tumor proliferation, tumor invasion, tumor density, vascularity, vascular permeability, microvascular density and metabolite profiles. Exploratory analyses will utilize quantitative imaging tumor metrics and radiome sequencing for texture maps to assess gene signatures of tumor cell apoptosis, invasion and immune cell infiltration. Exploratory analysis using quantitative imaging tumor metrics and texture maps will also be used to assess pseudoprogression, progression and response. These analyses will be compared to a retrospective cohort of patients that have been dichotomously analyzed for lack of inflammatory response versus robust intratumoral inflammatory responses to prospectively validate the sensitivity and specificity of this approach.

Product: MK-3475


79

Analysis results of Tumor-infiltrating lymphocytes will be summarized using descriptive statistics.

Patient responses to the select items of the PRO-CTCAE will be examined over time using descriptive statistics to capture the patient symptom toxicity.

Microbiome analyses will utilize (1) gene expression for a variety of genes in normal skin vs. skin area with rash for patients that experience dermatologic irAEs, (2) gene expression for a variety of genes at baseline, at onset of toxicity, and time of tumor restaging for patients that experience oral irAEs, and (3) gene expression for a variety of genes at baseline, at onset of toxicity, time of tumor restaging, and end of treatment visit for patients that experience gut irAEs. These analyses will explore differentially expressed genes between normal skin and skin with rash and will explore differentially expressed genes at onset of toxicity comparing to baseline for patients that experience oral irAEs and for patients that experience gut irAEs. The threshold of absolute fold change≥1.3 and Benjamini-Hochberg adjusted p<0.2 will be used to identify biologically meaningful sets of differentially expressed genes. <sup>18</sup> Due to exploratory nature of this analysis, we may use different significant criteria.

### 8.5.2 Analysis Populations

The population analysis will be evaluated as aggregate data, by tumor indication, and between PD-L1 and non-PD-L1 expressing tumor types.

### 8.5.2.1 Efficacy Analysis Populations

There will be 10 cohorts included in the overall population of different cancer types. The safety population will be the main population for all analyses (demographics, efficacy and safety) unless otherwise stated. The modified intent-to-treat (ITT) population will include all patients enrolled in the study that received at least one dose of drug.

#### 8.5.3 Statistical Methods

Tabulations will be produced for appropriate demographic, baseline, efficacy and safety parameters. For categorical variables, summary tabulations of the number and percentage of subjects within each category (with a category for missing data) of the parameter will be presented, as well as two-sided 95% confidence intervals, unless otherwise stated. For continuous variables, the number of subjects, mean, median, standard deviation (SD), minimum, and maximum values will be presented. Time-to-event data will be summarized using Kaplan-Meier methodology using 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals, as well as percentage of censored observations.

No imputation of missing efficacy data is planned. For time to event analyses, patients who have no efficacy evaluations for disease recurrence will be considered censored at time 0.

Product: MK-3475

Product: MK-3475 80 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

For adverse events (AEs), missing dates will not be imputed, however, if partial dates are available, they will be used to assess if the AE occurred during the treatment period. Missing severities of AEs will not be imputed and will be considered missing in any tabulations of AE severity. If an AE is missing a response to the question regarding relationship to treatment, the event will be considered to be related.

No adjustments for multiple testing will be performed. All inferences beyond those involved in the Simon design will be considered exploratory. Unless otherwise stated, all statistical tests will be conducted at the  $\alpha$ =0.05 (2-sided) level.

The statistical analysis of the data obtained from the PRO-CTCAE questionnaires will be performed. We will use primarily descriptive statistics to describe how patients rated symptoms over time. We will construct lowess curves for each symptom to graphically display how symptom changes over time.

# 9.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL SUPPLIES

### 9.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Clinical Supplies will be provided by Merck as summarized in Table 9.

**Table 9 Product Descriptions** 

| Product Name & Potency | Dosage Form |
|---------------------------|----------------------------------|
| Pembrolizumab 50 mg | Lyophilized Powder for Injection |
| Pembrolizumab 100 mg/ 4mL | Solution for Injection |

### 9.2 Packaging and Labeling Information

Clinical supplies will be affixed with a clinical label in accordance with regulatory requirements.

Product: MK-3475

81 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

#### 9.3 Clinical Supplies Disclosure

This trial is open-label; therefore, the subject, the trial site personnel, the IND Sponsor and/or designee are not blinded to treatment. Drug identity (name, strength) is included in the label text; random code/disclosure envelopes or lists are not provided.

### **Storage and Handling Requirements**

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

#### **Returns and Reconciliation**

The investigator is responsible for keeping accurate records of the clinical supplies received from Merck or designee, the amount dispensed to and returned by the subjects and the amount remaining at the conclusion of the trial.

Upon completion or termination of the study, all unused and/or partially used investigational product will be destroyed at the site per institutional policy. It is the Investigator's responsibility to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable federal, state, local and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

#### 10.0 ADMINISTRATIVE AND REGULATORY DETAILS

### 10.1 Confidentiality

### 10.1.1 Confidentiality of Data

By signing this protocol, the investigator affirms to the IND Sponsor that information furnished to the investigator by the IND Sponsor will be maintained in confidence, and such information will be divulged to the institutional review board, ethics review committee (IRB/ERC) or similar or expert committee; affiliated institution and employees, only under an appropriate understanding of confidentiality with such board or committee, affiliated institution and employees. Data generated by this trial will be considered confidential by the investigator, except to the extent that it is included in a publication as provided in the Publications section of this protocol.

Product: MK-3475

Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27.Jan2022

82

### 10.1.2 Confidentiality of Subject Records

By signing this protocol, the investigator agrees that the IND Sponsor (or Sponsor representative), IRB/ERC, or regulatory authority representatives may consult and/or copy trial documents in order to verify worksheet/case report form data. By signing the consent form, the subject agrees to this process. If trial documents will be photocopied during the process of verifying worksheet/case report form information, the subject will be identified by unique code only; full names/initials will be masked prior to transmission to the IND Sponsor.

By signing this protocol, the investigator agrees to treat all subject data used and disclosed in connection with this trial in accordance with all applicable privacy laws, rules and regulations.

### 10.1.3 Confidentiality of Investigator Information

By signing this protocol, the investigator recognizes that certain personal identifying information with respect to the investigator, and all subinvestigators and trial site personnel, may be used and disclosed for trial management purposes, as part of a regulatory submissions, and as required by law. This information may include:

- 1. Name, address, telephone number and e-mail address;
- 2. Hospital or clinic address and telephone number;
- 3. Curriculum vitae or other summary of qualifications and credentials; and
- 4. Other professional documentation.

Consistent with the purposes described above, this information may be transmitted to the IND Sponsor, and subsidiaries, affiliates and agents of the Merck, in your country and other countries, including countries that do not have laws protecting such information. Additionally, the investigator's name and business contact information may be included when reporting certain serious adverse events to regulatory authorities or to other investigators. By signing this protocol, the investigator expressly consents to these uses and disclosures.

If this is a multicenter trial, in order to facilitate contact between investigators, the IND Sponsor may share an investigator's name and contact information with other participating investigators upon request.

### 10.1.4 Data Sharing

Study data, imaging, and samples will not be shared with any individuals or entities unless specified in a clinical trial agreement or data or material transfer agreement.

Product: MK-3475

83 27Jan2022 Protocol/Amendment No.: Version 17/ MDACC#2015-0948

De-identified data, including, but not limited to tumor type, tumor response, and toxicity, and de-identified scans and imaging will be reviewed by the collaborator, Rivka Colen at University of Pittsburgh, to provide expertise in the statistical analyses for the relationship of immune cell metabolism and radiomics. A waiver of consent will be utilized for patients that cannot be reconsented. Results from the analysis will be sent to the PI.

De-identified data output from RNA sequencing performed on tumor samples will be reviewed by the collaborator, Daniel Lee, MD, PhD, at InSilico Genomics to provide expertise in the statistical analyses for the relationship of epigenetic signatures and provide a score for clinical outcomes and markers. No clinical data will be sent to Dr. Lee. All clinical data and epigenetics scoring will be correlated here at MDACC. A waiver of consent will be utilized for patients that cannot be reconsented.

De-identified data, including, but not limited to tumor type, tumor response, toxicity, translational data, and baseline plasma samples will be sent to the collaborator, Stephen Johnston, PhD at Arizona State University to perform HD peptide analyses. A waiver of consent will be utilized for patients that cannot be reconsented. Results from the analysis will be sent to the PI.

De-identified data, including, but not limited to personal hygiene, antibiotic use, medication use, tumor type, tumor response, and toxicity, and de-identified samples will be reviewed by the collaborator, Julia Oh, PhD at Jackson Laboratory to provide expertise in the skin, stool, and oral microbiome analyses for the relationship microbiome and immune-related toxicity. De-identified clinical data will be coded to the samples; however, the code will only be available to the PI and MDACC study team. A waiver of consent will be utilized for patients that cannot be reconsented. Results from the analysis will be sent to the PI.

De-identified data, including, but not limited to tumor type, tumor response, toxicity, translational data, and two (baseline and on-treatment) samples (plasma or serum) for up to 130 patients will be sent to the collaborator, Ronan McDaid, at Oncimmune to perform autoantibody profiling analyses. A waiver of consent will be utilized for patients that cannot be reconsented. Results from the analysis will be sent to the PI.

H&E stained whole slide images will be uploaded to the webpage of collaborator, Chan-Young Ock, MD, PhD at Lunit Inc. to analyze tumor-infiltrating lymphocytes. A waiver of consent will be utilized for patients that cannot be reconsented. Results from the analysis will be sent to the PI. Lunit SCOPE IO is an artificial intelligence (AI)-powered spatial tumor-infiltrating lymphocytes analyzer. Lunit SCOPE IO classifies Immune Phenotype (IP) of each region of interest (ROI) in the tumor microenvironment: inflamed immune phenotype as high TIL density within the cancer area; immune-excluded immune phenotype as high TIL density exclusively in the cancer stroma; immune-desert immune phenotype as low TIL density in both the cancer area and cancer stroma. The Inflamed Score (IS) or Immune-Excluded Score (IES) are defined as the proportion of all tumor-containing tiles within a WSI classified as being of the inflamed IP or immune-excluded IP. Lunit SCOPE IO will be accessed via a web interface for slide image analysis and return of results. H&E stained whole slide images will be uploaded

Product: MK-3475


84

to the webpage of collaborator, Chan-Young Ock, MD, PhD at Lunit Inc. to analyze tumor-infiltrating lymphocytes. A waiver of consent will be utilized for patients that cannot be reconsented. Results from the analysis will be sent to the PI.

Data sent outside of MDACC will not have identifying patient information included.

### 10.2 Compliance with Financial Disclosure Requirements

Financial Disclosure requirements are outlined in the US Food and Drug Administration Regulations, Financial Disclosure by Clinical Investigators (21 CFR Part 54). It is the IND Sponsor's responsibility to determine, based on these regulations, whether a request for Financial Disclosure information is required. It is the investigator's/subinvestigator's responsibility to comply with any such request.

The investigator/subinvestigator(s) agree, if requested by the IND Sponsor in accordance with 21 CFR Part 54, to provide his/her financial interests in and/or arrangements with the IND Sponsor to allow for the submission of complete and accurate certification and disclosure statements. The investigator/subinvestigator(s) further agree to provide this information on Certification/Disclosure Form, commonly known as a financial disclosure form, provided by the IND Sponsor or through a secure password-protected electronic portal provided by the IND Sponsor. The investigator/subinvestigator(s) also consent to the transmission of this information to the IND Sponsor in the United States for these purposes. This may involve the transmission of information to countries that do not have laws protecting personal data.

### 10.3 Compliance with Law, Audit and Debarment

By signing this protocol, the investigator agrees to conduct the trial in an efficient and diligent manner and in conformance with this protocol; generally accepted standards of Good Clinical Practice (e.g., International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice: Consolidated Guideline and other generally accepted standards of good clinical practice); and all applicable federal, state and local laws, rules and regulations relating to the conduct of the clinical trial.

The investigator also agrees to allow monitoring, audits, IRB/ERC review and regulatory authority inspection of trial-related documents and procedures and provide for direct access to all trial-related source data and documents.

The investigator agrees not to seek reimbursement from subjects, their insurance providers or from government programs for procedures included as part of the trial reimbursed to the investigator by the Sponsor.

The investigator shall prepare and maintain complete and accurate trial documentation in compliance with Good Clinical Practice standards and applicable federal, state and local

Product: MK-3475

85 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

laws, rules and regulations; and, for each subject participating in the trial, provide all data, and, upon completion or termination of the clinical trial, submit any other reports to the IND Sponsor as required by this protocol or as otherwise required pursuant to any agreement with the IND Sponsor.

Trial documentation will be promptly and fully disclosed to the IND Sponsor by the investigator upon request and also shall be made available at the trial site upon request for inspection, copying, review and audit at reasonable times by representatives of the IND Sponsor or any regulatory authorities. The investigator agrees to promptly take any reasonable steps that are requested by the IND Sponsor as a result of an audit to cure deficiencies in the trial documentation and worksheets/case report forms.

The investigator must maintain copies of all documentation and records relating to the conduct of the trial in compliance with all applicable legal and regulatory requirements. This documentation includes, but is not limited to, the protocol, worksheets/case report forms, advertising for subject participation, adverse event reports, subject source data, correspondence with regulatory authorities and IRBs/ERCs, consent forms, investigator's curricula vitae, monitor visit logs, laboratory reference ranges, laboratory certification or quality control procedures and laboratory director curriculum vitae. By signing this protocol, the investigator agrees that documentation shall be retained until at least 2 years after the last approval of a marketing application in an ICH region or until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. Because the clinical development and marketing application process is variable, it is anticipated that the retention period can be up to 15 years or longer after protocol database lock. The IND Sponsor will determine the minimum retention period and notify the investigator when documents may be destroyed. The IND Sponsor also recognizes that documents may need to be retained for a longer period if required by local regulatory requirements. All trial documents shall be made available if required by relevant regulatory authorities. The investigator must consult with and obtain written approval by the IND Sponsor prior to discarding trial and/or subject files.

ICH Good Clinical Practice guidelines recommend that the investigator inform the subject's primary physician about the subject's participation in the trial if the subject has a primary physician and if the subject agrees to the primary physician being informed.

The investigator will promptly inform the IND Sponsor of any regulatory authority inspection conducted for this trial.

Persons debarred from conducting or working on clinical trials by any court or regulatory authority will not be allowed to conduct or work on this IND Sponsor's trials. The investigator will immediately disclose in writing to the IND Sponsor if any person who is involved in conducting the trial is debarred or if any proceeding for debarment is pending or, to the best of the investigator's knowledge, threatened.

Product: MK-3475

86 27Jan2022 Protocol/Amendment No.: Version 17/ MDACC#2015-0948

In the event the IND Sponsor prematurely terminates a particular trial site, the IND Sponsor will promptly notify that trial site's IRB/IEC.

According to European legislation, a IND Sponsor must designate an overall coordinating investigator for a multi-center trial (including multinational). When more than one trial site is open in an EU country, Merck, as the IND Sponsor, will designate, per country, a national principal coordinator (Protocol CI), responsible for coordinating the work of the principal investigators at the different trial sites in that Member State, according to national regulations. For a single-center trial, the Protocol CI is the principal investigator. In addition, the IND Sponsor must designate a principal or coordinating investigator to review the trial report that summarizes the trial results and confirm that, to the best of his/her knowledge, the report accurately describes the conduct and results of the trial [Clinical Study Report (CSR) CI]. The IND Sponsor may consider one or more factors in the selection of the individual to serve as the Protocol CI and or CSR CI (e.g., availability of the CI during the anticipated review process, thorough understanding of clinical trial methods, appropriate enrollment of subject cohort, timely achievement of trial milestones). The Protocol CI must be a participating trial investigator.

### 10.4 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to the Clinical Trials Data Bank, http://www.clinicaltrials.gov. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

#### 10.5 Quality Management System

By signing this protocol, the IND Sponsor agrees to be responsible for implementing and maintaining a quality management system with written development procedures and functional area standard operating procedures (SOPs) to ensure that trials are conducted and data are generated, documented, and reported in compliance with the protocol, accepted standards of Good Clinical Practice, and all applicable federal, state, and local laws, rules and regulations relating to the conduct of the clinical trial.

### 10.6 Data Management

The investigator or qualified designee is responsible for recording and verifying the accuracy of subject data. By signing this protocol, the investigator acknowledges that his/her electronic signature is the legally binding equivalent of a written signature. By entering his/her electronic signature, the investigator confirms that all recorded data have

Product: MK-3475 87

been verified as accurate.

This study will be monitored by the University of Texas MD Anderson IND Office, and a protocol-specific monitoring plan will be followed.

All patients who meet eligibility criteria and are enrolled in this trial will be registered in Clinical Oncology Research Database (CORe) at the University of Texas MD Anderson Cancer Center at Houston. Data will be collected and stored in the Investigational Cancer Therapeutics database, Molecular and Clinical Data Integrated Platform (MOCLIP).

Product: MK-3475

88 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

### 11.0 APPENDICES

### 11.1 ECOG Performance Status

| Grade | Description |
|---|---|
| 0 | Normal activity. Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| 5 | Dead. |

<sup>\*</sup> As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982. The Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair.

Product: MK-3475
27Jan2022

### 11.2 Common Terminology Criteria for Adverse Events V4.03 (CTCAE)

The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html)

Product: MK-3475


90

### 11.3 Response Evaluation Criteria in Solid Tumors (RECIST)

RECIST version 1.1\* or irRECIST will be used in this study for assessment of tumor response. While either CT or MRI may be utilized, as per RECIST 1.1 or irRECIST, CT is the preferred imaging technique in this study.

\* As published in the European Journal of Cancer:

E.A. Eisenhauer, P. Therasse, J. Bogaerts, L.H. Schwartz, D. Sargent, R. Ford, J. Dancey, S. Arbuck, S. Gwyther, M. Mooney, L. Rubinstein, L. Shankar, L. Dodd, R. Kaplan, D. Lacombe, J. Verweij. New response evaluation criteria in solid tumors: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47.

Bohnsack O, Hoos A, Ludajic K. Adaptation of the immune related response criteria: irRECIST Ann Oncol 2014;25(suppl 4):11 Abstract 1070.

In addition, volumetric analysis will be explored by central review for response assessment.

Product: MK-3475

91 Protocol/Amendment No.: Version 17/ MDACC#2015-0948 27Jan2022

#### 12.0 REFERENCES

Eisenhauer EA, Therasse P, Bogaerts J, et al: New response evaluation criteria 1. in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer 45:228-47, 2009

- Corp. MSD: Pembrolizumab Investigator's Brochure, 2015
- 3. Disis ML: Immune regulation of cancer. J Clin Oncol 28:4531-8, 2010
- 4. Yang I, Tihan T, Han SJ, et al: CD8+ T-cell infiltrate in newly diagnosed glioblastoma is associated with long-term survival. J Clin Neurosci 17:1381-5, 2010
- Dong H, Strome SE, Salomao DR, et al: Tumor-associated B7-H1 promotes Tcell apoptosis: a potential mechanism of immune evasion. Nat Med 8:793-800, 2002
- Sharpe AH, Freeman GJ: The B7-CD28 superfamily. Nat Rev Immunol 2:116-26, 2002
- Blackburn SD, Crawford A, Shin H, et al: Tissue-specific differences in PD-1 and PD-L1 expression during chronic viral infection: implications for CD8 T-cell exhaustion. J Virol 84:2078-89, 2010
- Blank C, Brown I, Peterson AC, et al: PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res 64:1140-5, 2004
- 9. Bronte V, Mocellin S: Suppressive influences in the immune response to cancer. J Immunother 32:1-11, 2009
- Hodi FS, O'Day SJ, McDermott DF, et al: Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med 363:711-23, 2010
- Hamid O, Robert C, Daud A, et al: Safety and Tumor Responses with Lambrolizumab (Anti-PD-1) in Melanoma. New England Journal of Medicine 369:134-144, 2013
- 12. DiGiulio S: Keytruda Approved by FDA for Advanced Melanoma, Called 'Game Changer'. Oncology Times, 2014
- Francisco LM, Sage PT, Sharpe AH: The PD-1 pathway in tolerance and 13. autoimmunity. Immunol Rev 236:219-242, 2010
- Thompson RH, Dong H, Kwon ED: Implications of B7-H1 expression in clear cell carcinoma of the kidney for prognostication and therapy. Clinical cancer research 13:709s-715s, 2007
- Ohigashi Y, Sho M, Yamada Y, et al: Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clinical cancer research 11:2947-2953, 2005
- 16. McDermott DF, Atkins MB: PD-1 as a potential target in cancer therapy. Cancer medicine 2:662-673, 2013
- Simon R: Optimal two-stage designs for phase II clinical trials. Control Clin 17. Trials 10:1-10, 1989
- 18. Huggins CE, Domenighetti AA, Ritchie ME, et al: Functional and metabolic remodelling in GLUT4-deficient hearts confers hyper-responsiveness to substrate intervention. J Mol Cell Cardiol 44:270-80, 2008